CLINICAL TRIAL: NCT01976364
Title: A LONG-TERM, OPEN-LABEL EXTENSION STUDY OF TOFACITINIB (CP-690,550) FOR THE TREATMENT OF PSORIATIC ARTHRITIS
Brief Title: Open-Label Extension Study Of Tofacitinib In Psoriatic Arthritis
Acronym: OPAL BALANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3921092; 2011-002169-39 (EudraCT Number); OPAL BALANCE (Other: Alias Study Number)
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Results first posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Arthritis, Psoriatic
Keywords: Tofacitinib; Psoriatic Arthritis; Xeljanz; CP-690550; Jak-inhibitor; oral treatment; psoriasis; OPAL BALANCE; methotrexate; pruritus; itch; DLQI
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Pruritus | interventions — tofacitinib; Methotrexate

STUDY DESIGN:
Masking Description: The sub-study will be participant, care provider, investigator and outcomes assessor masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tofacitinib (Experimental)
  Interventions: Drug: Tofacitinib; Drug: Methotrexate; Drug: Placebo Methotrexate

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib 5 mg tablet twice daily
Drug: Tofacitinib — Tofactinib 10 mg tablet twice daily
Drug: Methotrexate — Methotrexate 7.5-20 mg weekly
  Other Names: Sub-study
Drug: Placebo Methotrexate — Placebo to match active methotrexate orally once a week
  Other Names: Sub-study

SUMMARY:
This is a Phase 3, long-term open-label extension study to evaluate the safety, tolerability and efficacy of tofacitinib in subjects with active PsA who have previously participated in randomized studies of tofacitinib for this indication.

This study will include a sub-study to evaluate the efficacy, safety and tolerability of tofacitinib 5 mg BID administered as monotherapy after methotrexate withdrawal compared to tofacitinib 5 mg BID continued in combination with methotrexate. The sub-study will be available to subjects who have completed at least 24 months of participation in the open-label extension study and meet eligibility criteria for the sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in qualifying PsA study involving tofacitinib

Exclusion Criteria:

* Time from End of Study visit of qualifying study is >3 months.
* Pregnant female, breastfeeding female or female of childbearing potential unwilling or unable to use highly effective birth control for duration of study and one ovulatory cycle thereafter.

Sub-study Inclusion Criteria:

* Subjects who have completed at least 24 months of treatment with tofacitinib in the extension study
* Subjects on a stable oral dose of methotrexate (maximum dose 20 mg per week)

Sub-study Exclusion Criteria:

-Subjects who are receiving methotrexate by a route other than oral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Actual)
Dates: Start 2014-02-17 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (152):
- United States (42):
  - Rheumatology Associates, PC, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Arizona Arthritis & Rheumatology Associates, P.C., Glendale, Arizona
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - Desert Medical Advances, Palm Desert, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Stanford Anatomic Pathology and Clinical Lab, Stanford, California
  - Stanford Health Care Department of Pharmacy lnvestigational Drug Services, Stanford, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - Rheumatology Associates of Central Florida, PA, Orlando, Florida
  - Millennium Research, Ormond Beach, Florida
  - Arthritis Center, Inc., Palm Harbour, Florida
  - Guillermo Valenzuela, MD PA dba Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - St. Luke's Clinic - Rheumatology, Boise, Idaho
  - St. Luke's Intermountain Research Center, Boise, Idaho
  - Bluegrass Community Research, Inc., Lexington, Kentucky
  - Klein and Associates, M.D., P.A., Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - St. Paul Rheumatology, P.A., Eagan, Minnesota
  - Clayton Medical Research, St Louis, Missouri
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cincinnati Rheumatic Disease Study Group, Inc., Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University Hospitals of Cleveland Medical Center, Cleveland, Ohio
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - East Penn Rheumatology Associates, PC, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Articularis Healthcare Group, Inc d/b/a Low Country Rheumatology, Summerville, South Carolina
  - Arthritis Clinic, Jackson, Tennessee
  - West Tennessee Research Institute, Jackson, Tennessee
  - Adriana Pop-Moody MD Clinic PA, Corpus Christi, Texas
  - Pioneer Research Solutions, Inc., Cypress, Texas
  - Investigational Drug Services, Salt Lake City, Utah
  - University of Utah Hospital & Clinics, Salt Lake City, Utah
  - University of Utah Hospitals and Clinics - Clinie 2, Salt Lake City, Utah
  - Swedish Medical Center, Seattle, Washington
  - Seattle Rheumatology Associates, Seattle, Washington
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Rheumatology Research Unit, Maroochydore, Queensland
  - Pacific Private Clinic, Southport, Queensland
  - Emeritus Research, Camberwell, Victoria
  - St. Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - St. Vincent's Hospital, Fitzroy, Victoria
- Belgium (6):
  - Hopital Erasme - Clinique Universitaire de Bruxelles, Brussels, Brabant Flamand
  - Hopital Erasme - Clinique Universitaire de Bruxelles, Brussels
  - Reumaclinic, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - University Hospital Leuven, Leuven
  - ZNA Jan Palfijn, Merksem
- Brazil (3):
  - CMIP- Centro Mineiro de Pesquisa Ltda/CETAL- Centro de Estudos e Tratamento do Aparelho Locomotor, Juiz de Fora, Minas Gerais
  - EDUMED - Educação em Saùde SS Ltda, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre (HCPA) / UFRGS, Porto Alegre, Rio Grande do Sul
- Bulgaria (4):
  - UMHAT "Dr. G. Stranski" EAD, Department of Rheumatology, Pleven
  - Multiprofile Hospital for Active Treatment - Plovdiv AD, Plovdiv
  - Multiprofile hospital for active treatment Kaspela EOOD, Plovdiv
  - Medical Center - "New rehabilitation center" EOOD, Stara Zagora
- K. Papp Clinical Research, Waterloo, Ontario, Canada
- Czechia (9):
  - X-Medica, s.r.o., Brno
  - Revmacentrum MUDr. Mostera, s.r.o., Brno
  - Stavovska, s.r.o., Brno
  - Revmatologie s.r.o., Brno
  - Vesalion s.r.o., Ostrava
  - Revmatologicky ustav - Lekarna, Prague
  - Revmatologicky ustav, Prague
  - Revmatologicka ambulance, Prague
  - MEDICAL PLUS, s.r.o., Uherské Hradiště
- Germany (10):
  - Rheumazentrum Prof. Dr. med Gunther Neeck, Bad Doberan, Mecklenburg-vorp
  - Charite Universitaetsmedizin Berlin, Berlin
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Rheumapraxis Steglitz, Berlin
  - Schlosspark-Klinik, Berlin
  - University Hospital of Cologne, Cologne
  - CIRI, Centrum fuer innovative Diagnostik und Therapie Rheumatologie und Immunologie (GmbH), Frankfurt am Main
  - Medizinische Universitaetsklinik Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Des Saarlandes Und Medizinische Fakultaet Der Universitaet Des Saarlandes, Homburg
  - Elisabeth Klinik Bigge, Olsberg
- Hungary (8):
  - Diagnoscan Magyarország Kft., Budapest
  - Budapest Fovaros II. keruleti Onkormanyzat Egeszsegugyi Szolgalata- Rontgen- Ultrahang, Budapest
  - Revita Reumatologiai Rendelo, Budapest
  - Qualiclinic Kft., Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont - Kozponti Radiologiai Diagnosztika Osztaly, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Reumatologiai Osztaly, Budapest
  - Csolnoky Ferenc Korhaz, Reumatologiai Osztaly, Veszprém
  - Csolnoky Ferenc Korhaz, Veszprém
- Mexico (12):
  - Hospital Angeles Clinica Londres, Mexico City, D.F
  - Centro Integral en Reumatologia S.A. de C.V., Guadalajara, Jalisco
  - Grupo Medico Camino S.C., Mexico City, Mexico City
  - Cliditer, S.A. DE C.V., Mexico City, Mexico City
  - Centro de Investigacion de Tratamientos Innovadores de Sinaloa, S.C., Culiacán, Sinaloa
  - Sanatorio CEMSI Chapultepec, Culiacán, Sinaloa
  - Hospital General de Culiacan Dr. Bernardo J. Gastelum, Culiacán, Sinaloa
  - Instituto Medico Panamericano, S.A de C.V., Mérida, Yucatán
  - Unidad Reumatologica Las Americas S.C.P., Mérida, Yucatán
  - Centro Multidisciplinario Para El Desarrollo Especializado De La Investigacion Clinica En, Mérida, Yucatán
  - Christus Muguerza del Parque S.A. de C.V., Chihuahua City
  - Investigacion y Biomedicina de Chihuahua SC, Chihuahua City
- Poland (19):
  - Centrum Medyczne Pratia S.A. Warszawa, Warsaw, Masovian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Przychodnia Chirurgiczna dla Dzieci "PriamaMed" Sp.P., Bialystok
  - Zdrowie Osteo-Medic s.c. L. i A. Racewicz, A. i J. Supronik, Bialystok
  - ClinicMed Daniluk, Nowak Spolka Jawna, Bialystok
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Kliniczno-Badawcze J.Brzezicki, B.Gornikiewicz-Brzezicka Lekarze Spolka partnerska, Elblag
  - Centrum Radiologii, Elblag
  - NZOZ Centrum Reumatologiczne Indywidualna Specjalistyczna Praktyka Lekarska Lek. Med. Barbara Bazela, Elblag
  - Wojewodzki Szpital Zespolony, Zaklad Radiologii, Elblag
  - Przychodnia Specjalistyczna Lekarskiej Spoldzielni Pracy "Medica", Grodzisk Mazowiecki
  - Specjalistyczne Gabinety Lekarskie "DERMED" Anna Kaszuba, Lodz
  - Zespol Poradni Specjalistycznych Reumed Filia Onyksowa, Lublin
  - Top-Medical Sp. z o. o., Lublin
  - NZOZ Lecznica MAK-MED s.c., Nadarzyn
  - Prywatna Praktyka Lekarska Prof. UM dr hab. med. Pawel Hrycaj, Poznan
  - NZOZ Nasz Lekarz Praktyka Grupowa Lekarzy Rodzinnych z Przychodnia Specjalistyczna w Toruniu, Torun
  - Rheuma-Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - Reumatika Centrum Reumatologii NZOZ, Warsaw
  - Synexus Polska Oddzial we Wroclawiu, Wroclaw
- Russia (9):
  - State Autonomic Healthcare Institution ''City Clinical Hospital # 7'', Kazan', Tatarstan Republic
  - SBIH of Moscow "City Clinical Hospital #1 n. a. N.I. Pirogov" of the Healthcare Department of Moscow, Moscow
  - Research Institution of Fundamental and Clinical Immunology, Novosibirsk
  - Limited Liability Company Consultative Diagnostic Rheumatology Center "Healthy Joints", Novosibirsk
  - Regional State Budgetary Health Care Institution of Karelia Republic, Petrozavodsk
  - State Institution of Healthcare Regional Clinical Hospital, Saratov
  - State Budget Educational Institution of Highest Professional Education, Tomsk
  - State Autonomous Healthcare lnstitution of Yaroslavl Region "Clinical Hospital of Emergency Medical, Yaroslavl
  - State Healthcare Institution of Yaroslavl Region Clinical Emergency Hospital n.a.N.V. Solovyev, Yaroslavl
- Slovakia (3):
  - Nestatna reumatologicka ambulancia, Bratislava
  - MEDMAN s.r.o. - reumatologicka ambulancia, Martin
  - REUMEX, s.r.o, Rimavská Sobota
- Spain (8):
  - Hospital Clinico de Santiago, Santiago de Compostela, A Coruna
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Complexo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Quiron Salud Infanta Luisa, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- Taiwan (4):
  - Buddhist Dalin Tzu Chi General Hospital, Chiayi City
  - Chang Gung Medical Foundation-Kaohsiung Branch, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (8):
  - Barking Havering and Redbridge University Hospital NHS Trust-King George Hospital, Goodmayes, Essex
  - Barking Havering and Redbridge University Hospitals NHS Trust, Romford, Essex
  - The Dudley Group NHS Foundation Trust, Dudley, WEST Midlands
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford, WEST Yorkshire
  - Bradford Royal lnfirmary, BTHFT, Bradford, WEST Yorkshire
  - Wirral University Teaching Hospital NHS Foundation Trust, Upton, Wirral
  - Royal United Hospitals NHS Foundation Trust, Bath
  - York Teaching Hospital NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Gossec L, Sellas A, Gruben DC, Valderrama M, Gomez S, Kinch C, Citera G. Response to Tofacitinib in Patients with Psoriatic Arthritis and Probable Anxiety/Depressive Disorder: A Post Hoc Analysis of Phase 3 Trials. Rheumatol Ther. 2025 Dec;12(6):1175-1186. doi: 10.1007/s40744-025-00800-7. Epub 2025 Oct 28. PMID 41148555
- [Derived] Gladman DD, Dougados M, Marzo-Ortega H, Cadatal MJ, Agarwal E, Kinch CD, Nash P. Long-term tofacitinib efficacy and safety in psoriatic arthritis with or without prior biologic DMARD exposure: a post hoc analysis. Rheumatol Adv Pract. 2025 Jan 21;9(2):rkaf008. doi: 10.1093/rap/rkaf008. eCollection 2025. PMID 40241921
- [Derived] Gladman DD, Nash P, Mease PJ, FitzGerald O, Duench S, Cadatal MJ, Masri KR. Efficacy and safety of tofacitinib in an open-label, long-term extension study in patients with psoriatic arthritis who received adalimumab or tofacitinib in a Phase 3 randomized controlled study: a post hoc analysis. Arthritis Res Ther. 2024 Dec 19;26(1):218. doi: 10.1186/s13075-024-03442-2. PMID 39702318
- [Derived] Nash P, Coates LC, Fleishaker D, Kivitz AJ, Mease PJ, Gladman DD, FitzGerald O, Wang C, Wu J, Hsu MA, Menon S, Fallon L, Kanik KS. Safety and efficacy of tofacitinib up to 48 months in patients with active psoriatic arthritis: final analysis of the OPAL Balance long-term extension study. Lancet Rheumatol. 2021 Apr;3(4):e270-e283. doi: 10.1016/S2665-9913(21)00010-2. Epub 2021 Mar 24. PMID 38279411
- [Derived] Nash P, Mease PJ, Fleishaker D, Wu J, Coates LC, Behrens F, Gladman DD, Kivitz AJ, Wei JC, Shirinsky I, Menon S, Romero AB, Fallon L, Hsu MA, Wang C, Kanik KS. Tofacitinib as monotherapy following methotrexate withdrawal in patients with psoriatic arthritis previously treated with open-label tofacitinib plus methotrexate: a randomised, placebo-controlled substudy of OPAL Balance. Lancet Rheumatol. 2021 Jan;3(1):e28-e39. doi: 10.1016/S2665-9913(20)30339-8. Epub 2020 Nov 16. PMID 38273637
- [Derived] Eder L, Gladman DD, Mease P, Pollock RA, Luna R, Aydin SZ, Ogdie A, Polachek A, Gruben D, Cadatal MJ, Kinch C, Strand V. Sex differences in the efficacy, safety and persistence of patients with psoriatic arthritis treated with tofacitinib: a post-hoc analysis of phase 3 trials and long-term extension. RMD Open. 2023 Mar;9(1):e002718. doi: 10.1136/rmdopen-2022-002718. PMID 36958766
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Nash P, Coates LC, Kivitz AJ, Mease PJ, Gladman DD, Covarrubias-Cobos JA, FitzGerald O, Fleishaker D, Wang C, Wu J, Hsu MA, Menon S, Fallon L, Romero AB, Kanik KS. Safety and Efficacy of Tofacitinib in Patients with Active Psoriatic Arthritis: Interim Analysis of OPAL Balance, an Open-Label, Long-Term Extension Study. Rheumatol Ther. 2020 Sep;7(3):553-580. doi: 10.1007/s40744-020-00209-4. Epub 2020 Jun 6. PMID 32506317
- [Derived] Burmester GR, Curtis JR, Yun H, FitzGerald O, Winthrop KL, Azevedo VF, Rigby WFC, Kanik KS, Wang C, Biswas P, Jones T, Palmetto N, Hendrikx T, Menon S, Rojo R. An Integrated Analysis of the Safety of Tofacitinib in Psoriatic Arthritis across Phase III and Long-Term Extension Studies with Comparison to Real-World Observational Data. Drug Saf. 2020 Apr;43(4):379-392. doi: 10.1007/s40264-020-00904-9. PMID 32006348
- [Derived] Gladman DD, Charles-Schoeman C, McInnes IB, Veale DJ, Thiers B, Nurmohamed M, Graham D, Wang C, Jones T, Wolk R, DeMasi R. Changes in Lipid Levels and Incidence of Cardiovascular Events Following Tofacitinib Treatment in Patients With Psoriatic Arthritis: A Pooled Analysis Across Phase III and Long-Term Extension Studies. Arthritis Care Res (Hoboken). 2019 Oct;71(10):1387-1395. doi: 10.1002/acr.23930. PMID 31112005
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921092&StudyName=Open-Label%20Extension%20Study%20Of%20Tofacitinib%20In%20Psoriatic%20Arthritis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants (who had previously participated in randomized psoriatic arthritis [PsA] clinical studies with tofacitinib) from qualifying studies A3921091 (NCT01877668) and A3921125 (NCT01882439) were enrolled into this current study A3921092 (NCT01976364).
Pre-assignment Details: This main study was a long-term extension study, which also included a sub-study (only for the purpose of efficacy, safety and tolerability of tofacitinib monotherapy as compared to tofacitinib combination therapy with methotrexate). Sub-study included eligible participants from main study who consented to take part in sub-study.
Groups:
- Tofacitinib: Participants with active psoriatic arthritis (PsA) received tofacitinib 5 milligram (mg) oral tablet, twice daily (BID) with or without allowed concomitant disease-modifying anti-rheumatic drugs (DMARDs) examples as methotrexate, leflunomide or sulfasalazine, as background therapy, for up to 36 months. Tofacitinib dose was increased to 10 mg BID or decreased back to 5 mg BID per investigator's discretion.
- Tofacitinib 5 mg BID + Methotrexate (MTX): Participants from main study received tofacitinib 5 mg oral tablet BID along with MTX capsules orally (dose range from 7.5 to 20 mg per week) for up to 12 months.
- Tofacitinib 5 mg BID + Placebo: Participants from main study received tofacitinib 5 mg oral tablet BID with MTX matched placebo capsules for up to 12 months.
Period: Main Study (36 Months)
Arm/Group | Tofacitinib | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Started | 686 | 0 | 0
Completed | 465 | 0 | 0
Not Completed | 221 | 0 | 0
Not completed — Adverse Event | 63 | 0 | 0
Not completed — Withdrawn due to pregnancy | 5 | 0 | 0
Not completed — Other | 13 | 0 | 0
Not completed — No longer met eligibility criteria | 2 | 0 | 0
Not completed — Medication error | 1 | 0 | 0
Not completed — Lost to Follow-up | 10 | 0 | 0
Not completed — Lack of Efficacy | 40 | 0 | 0
Not completed — Protocol Violation | 13 | 0 | 0
Not completed — Withdrawal by Subject | 69 | 0 | 0
Not completed — Death | 5 | 0 | 0
Period: Sub-study (12 Months)
Arm/Group | Tofacitinib | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Started | 0 | 89 (Participants from main study who consented to take part in sub-study, continued into sub-study.) | 90 (Participants from main study who consented to take part in sub-study, continued into sub-study.)
Completed | 0 | 83 | 85
Not Completed | 0 | 6 | 5
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Adverse Event | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants enrolled in this study who were part of a prior qualifying study, and who received at least one dose of open-label study medication in A3921092. Full analysis set (FAS) and the SAS were same in this study.
Groups:
- Tofacitinib: All Participants: All enrolled participants with PsA who were part of a prior qualifying study, and received at least one dose of open-label study medication (tofacitinib) in this study.
Arm/Group | Tofacitinib: All Participants
Number analyzed (Participants) | 686
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 370
  Male | 316
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 646
  More than one race | 17
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 48 months that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: Date of first dose of study medication up to 48 months (36 months of main study and 12 months of sub-study)
Population: SAS included all participants enrolled in this study who were part of a prior qualifying study, and who received at least one dose of open-label study medication in A3921092. Safety analysis included cumulative data for main and sub-study as pre-specified in protocol.
Measure: Number; unit: percentage of participants
Groups:
- All Participants: Main Study: Participants with active PsA received tofacitinib 5 mg oral tablet, BID with or without allowed concomitant DMARDs examples as methotrexate, leflunomide or sulfasalazine, as background therapy, for up to 36 months. Tofacitinib dose was increased to 10 mg BID or decreased back to 5 mg BID per investigator's discretion. Sub-study: Participants from main study received tofacitinib 5 mg oral tablet BID with MTX capsules orally (dose range from 7.5 to 20 mg per week) or tofacitinib 5 mg oral tablet BID with MTX matched placebo capsules, for up to 12 months.
Arm/Group | All Participants
Number analyzed (Participants) | 686
percentage of participants
  AEs | 83.7
  SAEs | 16.8

2. Primary Outcome: Number of Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs were classified into 3 categories according to their severity as mild AEs (did not interfere with participant's usual function), moderate AEs (interfered to some extent with participant's usual function) and severe AEs (interfered significantly with participant's usual function).
Time Frame: Date of first dose of study medication up to 48 months (36 months of main study and 12 months of sub-study)
Population: as for outcome 1
Measure: Number; unit: adverse events
Arm/Group | All Participants
Number analyzed (Participants) | 686
adverse events
  Number of adverse events: Mild | 1632
  Number of adverse events: Moderate | 1045
  Number of adverse events: Severe | 136

3. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Values
Description: Laboratory tests: hematology (Hb, hematocrit, RBC count, platelets, reticulocytes, WBC count, count and absolute lymphocytes,neutrophils, basophils, eosinophils, monocytes. Liver function (bilirubin [total, direct, indirect], AST, ALT, alkaline phosphatase, gamma-glutamyl transferase, albumin, total protein), renal function (blood urea nitrogen, creatinine), Lipids (cholesterol, HDL, LDL, triglyceride, apolipoprotein [A-1, B]), electrolytes (sodium, potassium, chloride, calcium, biocarbonate), chemistry (glucose, HbA1c, creatinine kinapse), urinalysis dipstick(urine pH, glucose, ketones, protein, blood, leukocyte, esterase), urinalysis microscopy (urine- RBC, WBC, bacteria, epithelial cells),C-reactive protein. Laboratory abnormality: determined by investigator per pre-defined criteria.
Time Frame: Date of first dose of study medication up to 48 months (36 months of main study and 12 months of sub-study)
Population: SAS included all participants enrolled in this study who were part of prior qualifying study, and who received at least 1 dose of open-label study medication in A3921092. Safety analysis include cumulative data for main and sub-study as pre-specified in protocol.Overall number of participants analyzed=participants evaluable for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 683
Participants | 646

4. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Values
Description: Laboratory tests: hematology (Hb, hematocrit, RBC count, platelets, reticulocytes, WBC count, count and absolute lymphocytes, neutrophils, basophils, eosinophils, monocytes. Liver function (bilirubin[total,direct,indirect], AST, ALT, alkaline phosphatase, gamma-glutamyl transferase, albumin, total protein), renal function (blood urea nitrogen, creatinine), Lipids(cholesterol, HDL, LDL, triglyceride, apolipoprotein [A-1, B]), electrolytes (sodium, potassium, chloride, calcium, biocarbonate), chemistry (glucose, HbA1c, creatinine kinapse), urinalysis dipstick(urine-pH, glucose, ketones, protein, blood, leukocyte, esterase), urinalysis microscopy(urine- RBC, WBC, bacteria, epithelial cells),C-reactive protein. Clinically significant change: determined by investigator per pre-defined criteria.
Time Frame: Date of first dose of study medication (Baseline) up to 48 months (36 months of main study and 12 months of sub-study)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 686
Participants | 9

5. Primary Outcome: Sub-study: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Month 6
Description: HAQ-DI assessed the degree of difficulty a participant had experienced during the past week in 8 domains of daily living activities: dressing/grooming, arising, eating, walking, reach, grip, hygiene, and other activities. There were total of 2-3 items distributed in each of these 8 domains. Each item was scored for level of difficulty on a 4-point scale from 0 to 3: 0= no difficulty; 1= some difficulty; 2= much difficulty; 3= unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible HAQ-DI score ranged from 0 (least difficulty) to 3 (extreme difficulty), where higher score indicated more difficulty while performing daily living activities.
Time Frame: Sub-study: Baseline (Day 1), Month 6
Population: FAS of sub-study included all participants who were randomized to the sub-study and received at least one dose of the sub-study drug (tofacitinib, MTX or placebo).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale | 0.0174 (0.02775) | 0.0428 (0.02714)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: Analysis was based on a repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline value; a common unstructured covariance matrix was used; Test type: Other; Least Squares (LS) Mean difference = 0.0255, 95% CI 2-sided [-0.0513 to 0.1022]

6. Primary Outcome: Sub-study: Change From Baseline in Psoriatic Arthritis Disease Activity Score (PASDAS) at Month 6
Description: PASDAS was composite PsA disease activity score that included following components: Physician and patient global assessment of disease activity (assessed on a 0-100 VAS) in millimeter (mm), swollen (66 joints) and tender joint counts (68 joints), Leeds enthesitis index (enthesitis assessed at 6 sites; total score of 0-6), tender dactylitic digit score (scored on a scale of 0-3, where 0= no tenderness and 3= extreme tenderness), short form-36 questionnaire (SF-36) physical component summary (norm-based domain scores were used in analyses; with a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity) and C-reactive protein (CRP) in milligram per liter (mg/L). PASDAS was composite score and was a weighted index with score range of 0 to 10, where higher score indicated more severe disease.
Time Frame: Sub-study: Baseline (Day 1), Month 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale | 0.138 (0.0805) | 0.229 (0.0786)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: Results were based on a repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline value; a common unstructured covariance matrix was used; Test type: Other; LS mean difference = 0.091, 95% CI 2-sided [-0.131 to 0.313]

7. Secondary Outcome: Main Study: Percentage of Participants Achieving an American College of Rheumatology 20 Percent (%) (ACR20) Response
Description: Participants with 20% improvement from baseline in tender and swollen joint counts and 20% improvement in at least 3 of the 5 measures: Patient's global assessment of arthritis (PtGA), Physician's global assessment of arthritis (PhyGA), participant's assessment of arthritis pain, HAQ-DI and C-reactive protein (CRP) in mg/L. PtGA: participant assessed health on VAS, 0 mm (very well) to 100 mm (worst health condition), higher score = worse condition. PhyGA: physician judged participants' pain on VAS, 0 (no pain) to 100 mm (extreme pain), higher score = more pain. Participant's assessment of arthritis pain: participant assessed pain on VAS, 0 mm (no pain) to 100 mm (most severe pain), higher score = more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score implied more disability.
Time Frame: Main Study: Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: FAS population for main study included all enrolled participants who were part of prior qualifying study, and who received at least 1 dose of tofacitinib in A3921092. Number analyzed=participants evaluable for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Tofacitinib: Participants with active PsA received tofacitinib 5 mg oral tablet, BID with or without allowed concomitant DMARDs examples as methotrexate, leflunomide or sulfasalazine, as background therapy, for up to 36 months. Tofacitinib dose was increased to 10 mg BID or decreased back to 5 mg BID per investigator's discretion.
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
percentage of participants
  Month 1: number analyzed (Participants) | 673
  Month 1 | 66.12 [62.55 to 69.70]
  Month 3: number analyzed (Participants) | 660
  Month 3 | 68.79 [65.25 to 72.32]
  Month 6: number analyzed (Participants) | 634
  Month 6 | 70.66 [67.12 to 74.21]
  Month 9: number analyzed (Participants) | 603
  Month 9 | 71.48 [67.87 to 75.08]
  Month 12: number analyzed (Participants) | 581
  Month 12 | 74.18 [70.62 to 77.74]
  Month 15: number analyzed (Participants) | 551
  Month 15 | 78.04 [74.58 to 81.50]
  Month 18: number analyzed (Participants) | 537
  Month 18 | 77.65 [74.13 to 81.18]
  Month 21: number analyzed (Participants) | 526
  Month 21 | 77.00 [73.40 to 80.59]
  Month 24: number analyzed (Participants) | 511
  Month 24 | 76.13 [72.43 to 79.82]
  Month 27: number analyzed (Participants) | 495
  Month 27 | 78.18 [74.54 to 81.82]
  Month 30: number analyzed (Participants) | 479
  Month 30 | 80.79 [77.27 to 84.32]
  Month 33: number analyzed (Participants) | 452
  Month 33 | 77.88 [74.05 to 81.70]
  Month 36: number analyzed (Participants) | 383
  Month 36 | 77.02 [72.81 to 81.24]

8. Secondary Outcome: Main Study: Percentage of Participants Achieving an American College of Rheumatology 50% (ACR50) Response
Description: Participants with 50% improvement from baseline in tender and swollen joint counts and 50% improvement in at least 3 of the 5 measures: PtGA, PhyGA, participant's assessment of arthritis pain, HAQ-DI and CRP in mg/L. PtGA: participant assessed health on VAS, 0 mm (very well) to 100 mm (worst health condition), higher score = worse condition. PhyGA: physician judged participants' pain on VAS, 0 (no pain) to 100 mm (extreme pain), higher score = more pain. Participant's assessment of arthritis pain: participant assessed pain on VAS, 0 mm (no pain) to 100 mm (most severe pain), higher score = more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score implied more disability.
Time Frame: Main Study: Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
percentage of participants
  Month 1: number analyzed (Participants) | 674
  Month 1 | 45.70 [41.94 to 49.46]
  Month 3: number analyzed (Participants) | 661
  Month 3 | 43.27 [39.49 to 47.04]
  Month 6: number analyzed (Participants) | 633
  Month 6 | 47.08 [43.19 to 50.97]
  Month 9: number analyzed (Participants) | 605
  Month 9 | 50.41 [46.43 to 54.40]
  Month 12: number analyzed (Participants) | 581
  Month 12 | 50.26 [46.19 to 54.32]
  Month 15: number analyzed (Participants) | 554
  Month 15 | 55.42 [51.28 to 59.55]
  Month 18: number analyzed (Participants) | 539
  Month 18 | 55.10 [50.90 to 59.30]
  Month 21: number analyzed (Participants) | 527
  Month 21 | 55.41 [51.16 to 59.65]
  Month 24: number analyzed (Participants) | 511
  Month 24 | 57.34 [53.05 to 61.63]
  Month 27: number analyzed (Participants) | 496
  Month 27 | 56.05 [51.68 to 60.42]
  Month 30: number analyzed (Participants) | 478
  Month 30 | 60.46 [56.08 to 64.84]
  Month 33: number analyzed (Participants) | 452
  Month 33 | 57.96 [53.41 to 62.52]
  Month 36: number analyzed (Participants) | 384
  Month 36 | 58.85 [53.93 to 63.78]

9. Secondary Outcome: Main Study: Percentage of Participants Achieving an American College of Rheumatology 70% (ACR70) Response
Description: Participants with 70% improvement from baseline in tender and swollen joint counts and 70% improvement in at least 3 of the 5 measures: PtGA, PhyGA, participant's assessment of arthritis pain, HAQ-DI and CRP in mg/L. PtGA: participant assessed health on VAS, 0 mm (very well) to 100 mm (worst health condition), higher score = worse condition. PhyGA: physician judged participants' pain on VAS, 0 (no pain) to 100 mm (extreme pain), higher score = more pain. Participant's assessment of arthritis pain: participant assessed pain on VAS, 0 mm (no pain) to 100 mm (most severe pain), higher score = more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score implied more disability.
Time Frame: Main Study: Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
percentage of participants
  Month 1: number analyzed (Participants) | 676
  Month 1 | 24.85 [21.59 to 28.11]
  Month 3: number analyzed (Participants) | 662
  Month 3 | 26.13 [22.79 to 29.48]
  Month 6: number analyzed (Participants) | 636
  Month 6 | 30.50 [26.92 to 34.08]
  Month 9: number analyzed (Participants) | 607
  Month 9 | 30.81 [27.13 to 34.48]
  Month 12: number analyzed (Participants) | 582
  Month 12 | 32.13 [28.34 to 35.92]
  Month 15: number analyzed (Participants) | 555
  Month 15 | 33.87 [29.94 to 37.81]
  Month 18: number analyzed (Participants) | 538
  Month 18 | 36.25 [32.18 to 40.31]
  Month 21: number analyzed (Participants) | 527
  Month 21 | 34.35 [30.29 to 38.40]
  Month 24: number analyzed (Participants) | 512
  Month 24 | 35.94 [31.78 to 40.09]
  Month 27: number analyzed (Participants) | 496
  Month 27 | 38.10 [33.83 to 42.38]
  Month 30: number analyzed (Participants) | 476
  Month 30 | 41.60 [37.17 to 46.02]
  Month 33: number analyzed (Participants) | 453
  Month 33 | 38.19 [33.72 to 42.66]
  Month 36: number analyzed (Participants) | 384
  Month 36 | 37.76 [32.91 to 42.61]

10. Secondary Outcome: Main Study: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Description: HAQ-DI assessed the degree of difficulty a participant had experienced during the past week in 8 domains of daily living activities: dressing/grooming, arising, eating, walking, reach, grip, hygiene, and other activities. There were total of 2-3 items distributed in each of these 8 domains. Each item was scored for level of difficulty on a 4-point scale from 0 to 3: 0= no difficulty; 1= some difficulty; 2= much difficulty; 3= unable to do. Overall score was computed as the sum of domain score and divided by the number of domains answered. Total possible HAQ-DI score range 0 (least difficulty) and 3 (extreme difficulty), where higher score indicated more difficulty while performing daily living activities.
Time Frame: Main Study: Baseline (Day 1), Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 675
  Change at Month 1 | -0.4373 (0.55677)
  Change at Month 3: number analyzed (Participants) | 661
  Change at Month 3 | -0.4559 (0.55104)
  Change at Month 6: number analyzed (Participants) | 636
  Change at Month 6 | -0.4755 (0.57468)
  Change at Month 9: number analyzed (Participants) | 605
  Change at Month 9 | -0.4841 (0.58294)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | -0.4782 (0.60163)
  Change at Month 15: number analyzed (Participants) | 554
  Change at Month 15 | -0.5108 (0.58277)
  Change at Month 18: number analyzed (Participants) | 539
  Change at Month 18 | -0.5116 (0.59401)
  Change at Month 21: number analyzed (Participants) | 528
  Change at Month 21 | -0.5211 (0.59568)
  Change at Month 24: number analyzed (Participants) | 511
  Change at Month 24 | -0.5068 (0.62016)
  Change at Month 27: number analyzed (Participants) | 496
  Change at Month 27 | -0.5219 (0.60833)
  Change at Month 30: number analyzed (Participants) | 478
  Change at Month 30 | -0.5356 (0.61316)
  Change at Month 33: number analyzed (Participants) | 453
  Change at Month 33 | -0.5276 (0.63803)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | -0.5476 (0.65226)

11. Secondary Outcome: Main Study: Percentage of Participants Achieving Psoriatic Arthritis Response Criteria (PsARC)
Description: PsARC is comprised of 4 clinical improvement criteria: greater than or equal to (>=) 20% improvement in PhyGA (VAS), >=20% improvement in PtGA; and >= 30% reduction in the number of tender joints; and >=30% reduction in the number of swollen joints. PtGA: participant assessed health on VAS, 0 mm (very well) to 100 mm (worst health condition), higher score = worse condition. PhyGA: physician judged participants' pain on VAS, 0 (no pain) to 100 mm (extreme pain), higher score = more pain. To achieve a clinical response, the participant must improve in 2 of the 4 PsARC criteria, 1 of which has to be the number of tender or swollen joints and none of the 4 score could worsen.
Time Frame: Main Study: Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
percentage of participants
  Month 1: number analyzed (Participants) | 669
  Month 1 | 68.46 [64.94 to 71.98]
  Month 3: number analyzed (Participants) | 657
  Month 3 | 69.56 [66.04 to 73.08]
  Month 6: number analyzed (Participants) | 633
  Month 6 | 73.14 [69.69 to 76.60]
  Month 9: number analyzed (Participants) | 599
  Month 9 | 74.46 [70.97 to 77.95]
  Month 12: number analyzed (Participants) | 577
  Month 12 | 76.08 [72.60 to 79.56]
  Month 15: number analyzed (Participants) | 547
  Month 15 | 79.52 [76.14 to 82.91]
  Month 18: number analyzed (Participants) | 534
  Month 18 | 80.15 [76.77 to 83.53]
  Month 21: number analyzed (Participants) | 522
  Month 21 | 79.50 [76.04 to 82.96]
  Month 24: number analyzed (Participants) | 507
  Month 24 | 77.51 [73.88 to 81.15]
  Month 27: number analyzed (Participants) | 494
  Month 27 | 80.16 [76.65 to 83.68]
  Month 30: number analyzed (Participants) | 475
  Month 30 | 82.11 [78.66 to 85.55]
  Month 33: number analyzed (Participants) | 449
  Month 33 | 80.85 [77.21 to 84.49]
  Month 36: number analyzed (Participants) | 381
  Month 36 | 77.17 [72.95 to 81.38]

12. Secondary Outcome: Main Study: Change From Baseline in Physician's Global Assessment of Psoriasis (PGA-PsO) Score (For Participants With Baseline PGA-PsO Score Greater Than [>]0) at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Description: The PGA-PsO was a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling were scored separately over the whole body according to a 5-point severity scale (0-4). Higher score indicated higher disease severity. Severity score for each erythema, induration and scaling were summed and averaged after which the total average was rounded to the nearest whole number score to determine a PGA-PsO score on a scale of 0 to 4 (0= clear, except for any residual discoloration, 1= almost clear, 2= mild, 3= moderate, 4= severe).
Time Frame: Main Study: Baseline (Day 1), Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: Analysis population included all enrolled participants who were part of a prior qualifying study, and who received at least one dose of tofacitinib in A3921092 and with baseline PGA-PsO score >0. Number analyzed =participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 660
units on a scale
  Change at Month 1: number analyzed (Participants) | 649
  Change at Month 1 | -1.1 (1.04)
  Change at Month 3: number analyzed (Participants) | 636
  Change at Month 3 | -1.1 (1.04)
  Change at Month 6: number analyzed (Participants) | 610
  Change at Month 6 | -1.2 (1.03)
  Change at Month 9: number analyzed (Participants) | 578
  Change at Month 9 | -1.2 (1.06)
  Change at Month 12: number analyzed (Participants) | 559
  Change at Month 12 | -1.1 (1.06)
  Change at Month 15: number analyzed (Participants) | 532
  Change at Month 15 | -1.2 (1.07)
  Change at Month 18: number analyzed (Participants) | 516
  Change at Month 18 | -1.2 (1.05)
  Change at Month 21: number analyzed (Participants) | 506
  Change at Month 21 | -1.2 (1.06)
  Change at Month 24: number analyzed (Participants) | 488
  Change at Month 24 | -1.3 (1.02)
  Change at Month 27: number analyzed (Participants) | 478
  Change at Month 27 | -1.3 (1.02)
  Change at Month 30: number analyzed (Participants) | 462
  Change at Month 30 | -1.3 (1.05)
  Change at Month 33: number analyzed (Participants) | 434
  Change at Month 33 | -1.3 (1.02)
  Change at Month 36: number analyzed (Participants) | 372
  Change at Month 36 | -1.2 (1.02)

13. Secondary Outcome: Main Study: Percentage of Participants With a Psoriasis Area and Severity Index 75 (PASI75) Score (For Participants With Baseline Body Surface Area [BSA]>=3% and Baseline PASI Score >0) at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Description: PASI: combined assessment of lesion severity and body area affected into single score; range =0 (no disease) -72 (maximal disease). Higher score representing greater severity of psoriasis. PASI is a composite scoring by investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk including axillae and groin, and lower limbs including buttocks). For each section % area of skin involved was estimated: 0 (0%) - 6 (90-100%) and severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1 =slight, 2 =moderate, 3 =marked, 4 =very marked. Final PASI =sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4). PASI75: at least a 75 % reduction in PASI relative to Baseline.
Time Frame: Main study: Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: Analysis population included all enrolled participants who were part of a prior qualifying study, and who received at least one dose of tofacitinib in A3921092 and with baseline BSA >=3% and baseline PASI score >0. Number analyzed =participants evaluable for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 474
percentage of participants
  Month 1: number analyzed (Participants) | 465
  Month 1 | 55.05 [50.53 to 59.58]
  Month 3: number analyzed (Participants) | 452
  Month 3 | 57.96 [53.41 to 62.52]
  Month 6: number analyzed (Participants) | 433
  Month 6 | 60.74 [56.14 to 65.34]
  Month 9: number analyzed (Participants) | 411
  Month 9 | 61.07 [56.36 to 65.78]
  Month 12: number analyzed (Participants) | 399
  Month 12 | 63.16 [58.42 to 67.89]
  Month 15: number analyzed (Participants) | 382
  Month 15 | 65.71 [60.95 to 70.47]
  Month 18: number analyzed (Participants) | 368
  Month 18 | 65.22 [60.35 to 70.08]
  Month 21: number analyzed (Participants) | 360
  Month 21 | 69.72 [64.98 to 74.47]
  Month 24: number analyzed (Participants) | 347
  Month 24 | 71.47 [66.72 to 76.22]
  Month 27: number analyzed (Participants) | 343
  Month 27 | 70.85 [66.04 to 75.66]
  Month 30: number analyzed (Participants) | 331
  Month 30 | 68.58 [63.58 to 73.58]
  Month 33: number analyzed (Participants) | 311
  Month 33 | 70.10 [65.01 to 75.18]
  Month 36: number analyzed (Participants) | 260
  Month 36 | 68.08 [62.41 to 73.74]

14. Secondary Outcome: Main Study: Percent Change From Baseline in PASI Composite Score (For Participants With Baseline BSA>=3% and Baseline PASI Score >0) at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Description: PASI: combined assessment of lesion severity & area affected into single score; range=0(no disease)-72(maximal disease). Higher score representing greater severity of psoriasis. PASI is a composite scoring by investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk including axillae and groin, and lower limbs including buttocks). For each section % area of skin involved was estimated: 0(0%) - 6(90-100%) & severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4).
Time Frame: Main study: Baseline, Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: Analysis population included all enrolled participants who were part of a prior qualifying study, and who received at least one dose of tofacitinib in A3921092 and with baseline BSA>=3% and baseline PASI score >0. Number analyzed =participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tofacitinib
Number analyzed (Participants) | 474
percent change
  At Month 1: number analyzed (Participants) | 465
  At Month 1 | -64.09 (57.473)
  At Month 3: number analyzed (Participants) | 452
  At Month 3 | -66.98 (43.647)
  At Month 6: number analyzed (Participants) | 433
  At Month 6 | -68.58 (44.568)
  At Month 9: number analyzed (Participants) | 411
  At Month 9 | -70.42 (40.617)
  At Month 12: number analyzed (Participants) | 399
  At Month 12 | -71.58 (42.515)
  At Month 15: number analyzed (Participants) | 382
  At Month 15 | -73.13 (43.653)
  At Month 18: number analyzed (Participants) | 368
  At Month 18 | -73.51 (40.527)
  At Month 21: number analyzed (Participants) | 360
  At Month 21 | -75.15 (44.182)
  At Month 24: number analyzed (Participants) | 347
  At Month 24 | -78.36 (34.808)
  At Month 27: number analyzed (Participants) | 343
  At Month 27 | -78.37 (34.405)
  At Month 30: number analyzed (Participants) | 331
  At Month 30 | -78.28 (30.270)
  At Month 33: number analyzed (Participants) | 311
  At Month 33 | -77.47 (43.952)
  At Month 36: number analyzed (Participants) | 260
  At Month 36 | -76.85 (31.973)

15. Secondary Outcome: Main Study: Percent Change From Baseline in PASI Clinical Signs Component Score (For Participants With Baseline BSA>=3% and Baseline PASI Score >0) at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Description: PASI: combined assessment of lesion severity & area affected into single score; range=0(no disease)-72(maximal disease). Higher score representing greater severity of psoriasis. PASI is a composite scoring by investigator of degree of clinical sign components for erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk including axillae and groin, and lower limbs including buttocks). For each section % area of skin involved was estimated: 0(0%) - 6(90-100%) and severity estimated by clinical signs components for erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4).
Time Frame: Main study: Baseline(Day 1), Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tofacitinib
Number analyzed (Participants) | 474
percent change
  Induration: At Month 1: number analyzed (Participants) | 456
  Induration: At Month 1 | -62.60 (62.288)
  Induration: At Month 3: number analyzed (Participants) | 442
  Induration: At Month 3 | -66.92 (46.898)
  Induration: At Month 6: number analyzed (Participants) | 423
  Induration: At Month 6 | -68.63 (46.644)
  Induration: At Month 9: number analyzed (Participants) | 402
  Induration: At Month 9 | -70.33 (41.960)
  Induration: At Month 12: number analyzed (Participants) | 390
  Induration: At Month 12 | -70.81 (48.439)
  Induration: At Month 15: number analyzed (Participants) | 373
  Induration: At Month 15 | -72.49 (48.644)
  Induration: At Month 18: number analyzed (Participants) | 359
  Induration: At Month 18 | -73.16 (40.801)
  Induration: At Month 21: number analyzed (Participants) | 352
  Induration: At Month 21 | -74.34 (47.617)
  Induration: At Month 24: number analyzed (Participants) | 338
  Induration: At Month 24 | -78.45 (36.534)
  Induration: At Month 27: number analyzed (Participants) | 335
  Induration: At Month 27 | -77.85 (34.297)
  Induration: At Month 30: number analyzed (Participants) | 322
  Induration: At Month 30 | -78.55 (31.187)
  Induration: At Month 33: number analyzed (Participants) | 303
  Induration: At Month 33 | -77.09 (42.305)
  Induration: At Month 36: number analyzed (Participants) | 256
  Induration: At Month 36 | -76.11 (35.000)
  Erythema: At Month 1: number analyzed (Participants) | 464
  Erythema: At Month 1 | -63.60 (67.818)
  Erythema: At Month 3: number analyzed (Participants) | 451
  Erythema: At Month 3 | -66.69 (43.013)
  Erythema: At Month 6: number analyzed (Participants) | 432
  Erythema: At Month 6 | -67.17 (46.756)
  Erythema: At Month 9: number analyzed (Participants) | 410
  Erythema: At Month 9 | -69.75 (42.882)
  Erythema: At Month 12: number analyzed (Participants) | 398
  Erythema: At Month 12 | -70.45 (46.575)
  Erythema: At Month 15: number analyzed (Participants) | 381
  Erythema: At Month 15 | -71.55 (50.406)
  Erythema: At Month 18: number analyzed (Participants) | 367
  Erythema: At Month 18 | -73.12 (45.194)
  Erythema: At Month 21: number analyzed (Participants) | 359
  Erythema: At Month 21 | -75.06 (45.993)
  Erythema: At Month 24: number analyzed (Participants) | 346
  Erythema: At Month 24 | -77.40 (38.093)
  Erythema: At Month 27: number analyzed (Participants) | 342
  Erythema: At Month 27 | -77.83 (33.877)
  Erythema: At Month 30: number analyzed (Participants) | 330
  Erythema: At Month 30 | -77.04 (33.478)
  Erythema: At Month 33: number analyzed (Participants) | 310
  Erythema: At Month 33 | -75.17 (53.782)
  Erythema: At Month 36: number analyzed (Participants) | 259
  Erythema: At Month 36 | -75.72 (34.823)
  Scaling: At Month 1: number analyzed (Participants) | 453
  Scaling: At Month 1 | -64.26 (55.848)
  Scaling: At Month 3: number analyzed (Participants) | 439
  Scaling: At Month 3 | -66.15 (52.568)
  Scaling: At Month 6: number analyzed (Participants) | 420
  Scaling: At Month 6 | -68.66 (49.145)
  Scaling: At Month 9: number analyzed (Participants) | 399
  Scaling: At Month 9 | -69.09 (48.506)
  Scaling: At Month 12: number analyzed (Participants) | 387
  Scaling: At Month 12 | -72.48 (45.755)
  Scaling: At Month 15: number analyzed (Participants) | 370
  Scaling: At Month 15 | -73.83 (42.528)
  Scaling: At Month 18: number analyzed (Participants) | 356
  Scaling: At Month 18 | -74.62 (39.708)
  Scaling: At Month 21: number analyzed (Participants) | 348
  Scaling: At Month 21 | -75.11 (44.570)
  Scaling: At Month 24: number analyzed (Participants) | 336
  Scaling: At Month 24 | -77.86 (38.041)
  Scaling: At Month 27: number analyzed (Participants) | 332
  Scaling: At Month 27 | -79.34 (31.825)
  Scaling: At Month 30: number analyzed (Participants) | 322
  Scaling: At Month 30 | -77.23 (37.819)
  Scaling: At Month 33: number analyzed (Participants) | 302
  Scaling: At Month 33 | -77.94 (41.688)
  Scaling: At Month 36: number analyzed (Participants) | 253
  Scaling: At Month 36 | -78.10 (30.391)

16. Secondary Outcome: Main Study: Change From Baseline in Dactylitis Severity Score (DSS) (For Participants With Baseline DSS Greater Than [>] 0) at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Description: Dactylitis was characterized by swelling of the entire finger or toe. The DSS was a function of finger circumference and tenderness, assessed and summed across all dactylitic digits. The severity of dactylitis was scored on a scale of 0-3, where 0 =no tenderness and 3 =extreme tenderness in each digit of the hands and feet. The range of total dactylitis severity score for a participant was 0-60. Higher score indicated greater severity.
Time Frame: Main study: Baseline (Day 1), Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: Analysis population included all enrolled participants who were part of a prior qualifying study, and who received at least one dose of tofacitinib in A3921092 and with baseline DSS >0. Number analyzed =participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 366
units on a scale
  Change at Month 1: number analyzed (Participants) | 360
  Change at Month 1 | -6.7 (7.65)
  Change at Month 3: number analyzed (Participants) | 352
  Change at Month 3 | -6.8 (7.71)
  Change at Month 6: number analyzed (Participants) | 335
  Change at Month 6 | -7.2 (7.89)
  Change at Month 9: number analyzed (Participants) | 313
  Change at Month 9 | -7.4 (7.29)
  Change at Month 12: number analyzed (Participants) | 305
  Change at Month 12 | -7.6 (7.70)
  Change at Month 15: number analyzed (Participants) | 290
  Change at Month 15 | -7.7 (7.44)
  Change at Month 18: number analyzed (Participants) | 282
  Change at Month 18 | -7.7 (7.50)
  Change at Month 21: number analyzed (Participants) | 275
  Change at Month 21 | -7.8 (7.89)
  Change at Month 24: number analyzed (Participants) | 269
  Change at Month 24 | -7.9 (7.76)
  Change at Month 27: number analyzed (Participants) | 265
  Change at Month 27 | -8.1 (7.59)
  Change at Month 30: number analyzed (Participants) | 257
  Change at Month 30 | -8.0 (7.65)
  Change at Month 33: number analyzed (Participants) | 250
  Change at Month 33 | -8.1 (7.75)
  Change at Month 36: number analyzed (Participants) | 212
  Change at Month 36 | -7.7 (7.88)

17. Secondary Outcome: Main Study: Change From Baseline in Leeds Enthesitis Index (LEI) (For Participants With Baseline LEI >0) at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Description: Enthesitis was inflammation in the tendon, ligament, and joint capsule fiber insertion into bone. The LEI assessed enthesitis in 6 sites including (right and left): lateral epicondyle humerus, medial femoral condyle and achilles tendon insertion. Tenderness is recorded as either present (score 1) or absent (score 0) for each of the 6 sites for a total score of 0-6. Higher score indicated a greater number of sites that are affected by enthesitis.
Time Frame: Main Study: Baseline (Day 1), Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: Analysis population included all enrolled participants who were part of a prior qualifying study, and who received at least one dose of tofacitinib in A3921092 and with baseline LEI >0. Number analyzed =participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 458
units on a scale
  Change at Month 1: number analyzed (Participants) | 449
  Change at Month 1 | -1.5 (1.88)
  Change at Month 3: number analyzed (Participants) | 437
  Change at Month 3 | -1.6 (1.79)
  Change at Month 6: number analyzed (Participants) | 418
  Change at Month 6 | -1.7 (1.78)
  Change at Month 9: number analyzed (Participants) | 398
  Change at Month 9 | -1.8 (1.80)
  Change at Month 12: number analyzed (Participants) | 380
  Change at Month 12 | -1.7 (1.82)
  Change at Month 15: number analyzed (Participants) | 364
  Change at Month 15 | -2.0 (1.76)
  Change at Month 18: number analyzed (Participants) | 347
  Change at Month 18 | -1.9 (1.79)
  Change at Month 21: number analyzed (Participants) | 340
  Change at Month 21 | -1.9 (1.81)
  Change at Month 24: number analyzed (Participants) | 327
  Change at Month 24 | -2.0 (1.72)
  Change at Month 27: number analyzed (Participants) | 317
  Change at Month 27 | -2.0 (1.73)
  Change at Month 30: number analyzed (Participants) | 306
  Change at Month 30 | -2.0 (1.76)
  Change at Month 33: number analyzed (Participants) | 288
  Change at Month 33 | -2.0 (1.75)
  Change at Month 36: number analyzed (Participants) | 253
  Change at Month 36 | -2.1 (1.76)

18. Secondary Outcome: Main Study: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index (For Participants With Baseline SPARCC Enthesitis Index >0) at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Description: The SPARCC enthesitis index identifies the presence or absence of tenderness at 16 enthesial sites, including (right and left): medial epicondyle humerus, lateral epicondyle humerus, supraspinatus insertion into greater tuberosity of humerus, greater trochanter, quadriceps insertion into superior border of patella, patellar ligament insertion into inferior pole of patella or tibial tubercle, Achilles tendon insertion into calcaneum and plantar fascia insertion into calcaneum. On examination, tenderness was recorded as present (1) or absent (0) for each of the 16 sites, with an overall total score ranging from 0 to 16. Higher score indicated a greater number of sites that are affected by enthesitis.
Time Frame: Main Study: Baseline (Day 1), Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: Analysis population included all enrolled participants who were part of a prior qualifying study, and who received at least one dose of tofacitinib in A3921092 and with baseline SPARCC enthesitis index >0. Number analyzed =participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 525
units on a scale
  Change at Month 1: number analyzed (Participants) | 517
  Change at Month 1 | -2.8 (3.60)
  Change at Month 3: number analyzed (Participants) | 504
  Change at Month 3 | -3.0 (3.61)
  Change at Month 6: number analyzed (Participants) | 481
  Change at Month 6 | -3.2 (3.72)
  Change at Month 9: number analyzed (Participants) | 457
  Change at Month 9 | -3.4 (3.69)
  Change at Month 12: number analyzed (Participants) | 438
  Change at Month 12 | -3.5 (3.46)
  Change at Month 15: number analyzed (Participants) | 415
  Change at Month 15 | -3.7 (3.55)
  Change at Month 18: number analyzed (Participants) | 400
  Change at Month 18 | -3.5 (3.45)
  Change at Month 21: number analyzed (Participants) | 394
  Change at Month 21 | -3.6 (3.60)
  Change at Month 24: number analyzed (Participants) | 379
  Change at Month 24 | -3.7 (3.62)
  Change at Month 27: number analyzed (Participants) | 369
  Change at Month 27 | -3.7 (3.56)
  Change at Month 30: number analyzed (Participants) | 359
  Change at Month 30 | -3.8 (3.49)
  Change at Month 33: number analyzed (Participants) | 340
  Change at Month 33 | -3.9 (3.39)
  Change at Month 36: number analyzed (Participants) | 290
  Change at Month 36 | -3.9 (3.69)

19. Secondary Outcome: Main Study: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score (For Participants With Presence of Spondylitis at Screening and Baseline BASDAI Score >0 cm) at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Description: BASDAI was a validated self-assessment tool used to determine disease activity in participants with ankylosing spondylitis. Utilizing a VAS of 0-10 cm (0= none and 10= very severe) participants answered 6 questions pertaining to 5 symptoms including fatigue, spinal pain, joint pain/swelling, areas of localized tenderness and morning stiffness. The final BASDAI score was an average of answers to 6 questions, with an overall possible score range of 0 to 10 centimeter (cm) with higher score represented more severe ankylosing spondylitis disease activity.
Time Frame: Main study: Baseline (Day 1), Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: Analysis population included all enrolled participants who were part of a prior qualifying study, and who received at least one dose of tofacitinib in A3921092 with presence of spondylitis at screening and baseline BASDAI Score>0 cm. Number analyzed =participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Tofacitinib
Number analyzed (Participants) | 124
centimeter
  Change at Month 1 | -2.26 (2.367)
  Change at Month 3: number analyzed (Participants) | 121
  Change at Month 3 | -2.10 (2.278)
  Change at Month 6: number analyzed (Participants) | 116
  Change at Month 6 | -2.40 (2.371)
  Change at Month 9: number analyzed (Participants) | 106
  Change at Month 9 | -2.35 (2.254)
  Change at Month 12: number analyzed (Participants) | 105
  Change at Month 12 | -2.41 (2.371)
  Change at Month 15: number analyzed (Participants) | 99
  Change at Month 15 | -2.35 (2.547)
  Change at Month 18: number analyzed (Participants) | 95
  Change at Month 18 | -2.41 (2.640)
  Change at Month 21: number analyzed (Participants) | 89
  Change at Month 21 | -2.28 (2.582)
  Change at Month 24: number analyzed (Participants) | 85
  Change at Month 24 | -2.47 (2.640)
  Change at Month 27: number analyzed (Participants) | 83
  Change at Month 27 | -2.65 (2.658)
  Change at Month 30: number analyzed (Participants) | 82
  Change at Month 30 | -2.95 (2.672)
  Change at Month 33: number analyzed (Participants) | 80
  Change at Month 33 | -2.85 (2.671)
  Change at Month 36: number analyzed (Participants) | 71
  Change at Month 36 | -2.88 (2.521)

20. Secondary Outcome: Main Study: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score (For Participants With Presence of Spondylitis at Screening and Baseline BASDAI Score >=4 cm) at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Description: BASDAI was a validated self-assessment tool used to determine disease activity in participants with ankylosing spondylitis. Utilizing a VAS of 0-10 cm (0= none and 10= very severe) participants answered 6 questions pertaining to 5 symptoms including fatigue, spinal pain, joint pain/swelling, areas of localized tenderness and morning stiffness. The final BASDAI score was an average of answers to 6 questions, with an overall possible score range of 0 to 10 cm with higher score represented more severe ankylosing spondylitis disease activity.
Time Frame: Main Study: Baseline (Day 1), Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36
Population: Analysis population included all enrolled participants who were part of a prior qualifying study, and who received at least one dose of tofacitinib in A3921092 and with presence of spondylitis at screening and baseline BASDAI score >=4 cm. Number analyzed =participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Tofacitinib
Number analyzed (Participants) | 106
centimeter
  Change at Month 1 | -2.59 (2.324)
  Change at Month 3: number analyzed (Participants) | 103
  Change at Month 3 | -2.41 (2.227)
  Change at Month 6: number analyzed (Participants) | 98
  Change at Month 6 | -2.74 (2.350)
  Change at Month 9: number analyzed (Participants) | 93
  Change at Month 9 | -2.63 (2.175)
  Change at Month 12: number analyzed (Participants) | 92
  Change at Month 12 | -2.65 (2.364)
  Change at Month 15: number analyzed (Participants) | 87
  Change at Month 15 | -2.65 (2.487)
  Change at Month 18: number analyzed (Participants) | 84
  Change at Month 18 | -2.65 (2.652)
  Change at Month 21: number analyzed (Participants) | 80
  Change at Month 21 | -2.47 (2.602)
  Change at Month 24: number analyzed (Participants) | 76
  Change at Month 24 | -2.72 (2.616)
  Change at Month 27: number analyzed (Participants) | 74
  Change at Month 27 | -2.90 (2.640)
  Change at Month 30: number analyzed (Participants) | 73
  Change at Month 30 | -3.27 (2.596)
  Change at Month 33: number analyzed (Participants) | 71
  Change at Month 33 | -3.17 (2.589)
  Change at Month 36: number analyzed (Participants) | 65
  Change at Month 36 | -3.08 (2.459)

21. Secondary Outcome: Main Study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Physical Component Summary Score at Months 1, 6, 12, 18, 24, 30 and 36
Description: The SF-36v2 acute was a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The 8 health domains were aggregated into two summary scores known as the physical component summary (PCS) score and the mental component summary (MCS) score. Norm-based domain scores, PCS and MCS scores were used in the analyses; each of which has a population mean of 50 with a standard deviation (SD) of 10 points, and ranges from minus infinity to plus infinity. A higher PCS score represented better physical health status.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: FAS of main study included all enrolled participants who were part of a prior qualifying study, and who received at least one dose of tofacitinib in A3921092. Number analyzed =participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 668
  Change at Month 1 | 6.44 (8.285)
  Change at Month 6: number analyzed (Participants) | 630
  Change at Month 6 | 6.71 (8.496)
  Change at Month 12: number analyzed (Participants) | 578
  Change at Month 12 | 7.23 (8.257)
  Change at Month 18: number analyzed (Participants) | 534
  Change at Month 18 | 7.44 (8.729)
  Change at Month 24: number analyzed (Participants) | 502
  Change at Month 24 | 7.79 (9.055)
  Change at Month 30: number analyzed (Participants) | 471
  Change at Month 30 | 8.06 (8.899)
  Change at Month 36: number analyzed (Participants) | 384
  Change at Month 36 | 7.77 (9.074)

22. Secondary Outcome: Main Study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Mental Component Summary Score at Months 1, 6, 12, 18, 24, 30, and 36
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The 8 health domains are aggregated into two summary scores known as the PCS score and the MCS score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher MCS score represents better mental health status.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 668
  Change at Month 1 | 4.72 (10.480)
  Change at Month 6: number analyzed (Participants) | 630
  Change at Month 6 | 4.98 (11.052)
  Change at Month 12: number analyzed (Participants) | 578
  Change at Month 12 | 5.25 (11.072)
  Change at Month 18: number analyzed (Participants) | 534
  Change at Month 18 | 5.53 (11.055)
  Change at Month 24: number analyzed (Participants) | 502
  Change at Month 24 | 5.79 (11.122)
  Change at Month 30: number analyzed (Participants) | 471
  Change at Month 30 | 5.82 (11.726)
  Change at Month 36: number analyzed (Participants) | 384
  Change at Month 36 | 6.18 (11.284)

23. Secondary Outcome: Main Study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Physical Functioning Domain Score at Months 1, 6, 12, 18, 24, 30, and 36
Description: SF-36v2 was a 36-item measure evaluating 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The 10 items of the physical functioning scale represented levels and kinds of limitations between extremes of physical activities, including lifting and carrying groceries; climbing stairs; bending, kneeling, or stooping; walking moderate distances; self-care limitations. The physical functioning items capture the presence and extent of physical limitations using a 3-level response continuum. Norm-based domain scores were used in the analyses; each of which had a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher physical functioning domain score represented better physical functioning.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | 6.06 (9.425)
  Change at Month 6: number analyzed (Participants) | 635
  Change at Month 6 | 6.44 (9.834)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | 7.00 (9.472)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | 7.31 (9.891)
  Change at Month 24: number analyzed (Participants) | 505
  Change at Month 24 | 7.69 (10.280)
  Change at Month 30: number analyzed (Participants) | 472
  Change at Month 30 | 7.96 (10.146)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | 7.80 (10.703)

24. Secondary Outcome: Main Study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Role-Physical Domain Score at Months 1, 6, 12, 18, 24, 30, and 36
Description: SF-36v2 acute was a 36-item measure evaluating 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health. The 4-item role-physical scale covers an array of physical health-related role limitations, including: a) limitations in the kind of work or other usual activities; b) reductions in the amount of time spent on work or other usual activities; c) difficulty performing work or other usual activities; & d) accomplishing less. Norm-based domain scores were used in the analyses; each of which had a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher role-physical domain score represented better role-physical functioning.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 669
  Change at Month 1 | 6.19 (9.545)
  Change at Month 6: number analyzed (Participants) | 631
  Change at Month 6 | 6.56 (9.650)
  Change at Month 12: number analyzed (Participants) | 579
  Change at Month 12 | 6.61 (9.293)
  Change at Month 18: number analyzed (Participants) | 534
  Change at Month 18 | 7.07 (10.050)
  Change at Month 24: number analyzed (Participants) | 503
  Change at Month 24 | 7.46 (10.094)
  Change at Month 30: number analyzed (Participants) | 473
  Change at Month 30 | 7.64 (10.041)
  Change at Month 36: number analyzed (Participants) | 384
  Change at Month 36 | 7.40 (9.996)

25. Secondary Outcome: Main Study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Bodily Pain Domain Score at Months 1, 6, 12, 18, 24, 30, and 36
Description: The SF-36v2 acute was a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The bodily pain scale comprises of 2 items pertaining to the intensity of bodily pain and extent of interference with normal work activities. Norm-based domain scores were used in the analyses; each of which had a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher bodily pain domain score represented less bodily pain.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 673
  Change at Month 1 | 8.36 (9.797)
  Change at Month 6: number analyzed (Participants) | 636
  Change at Month 6 | 8.52 (10.033)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | 9.29 (9.777)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | 9.70 (10.271)
  Change at Month 24: number analyzed (Participants) | 504
  Change at Month 24 | 9.95 (10.980)
  Change at Month 30: number analyzed (Participants) | 473
  Change at Month 30 | 10.21 (10.645)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | 10.45 (10.627)

26. Secondary Outcome: Main Study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) General Health Domain Score at Months 1, 6, 12, 18, 24, 30, and 36
Description: The SF-36v2 acute was a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The general health scale consisted of 5 items including a rating of health and 4 items addressing the respondent's view and expectations of his or her health. Norm-based domain scores were used in the analyses; each of which had a population mean of 50 with a SD of 10 points, and ranged from minus infinity to plus infinity. A higher general health domain score represented better general health perceptions.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | 3.89 (8.033)
  Change at Month 6: number analyzed (Participants) | 636
  Change at Month 6 | 4.09 (8.640)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | 4.68 (8.652)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | 4.76 (8.386)
  Change at Month 24: number analyzed (Participants) | 504
  Change at Month 24 | 4.89 (8.608)
  Change at Month 30: number analyzed (Participants) | 473
  Change at Month 30 | 4.81 (8.590)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | 4.36 (8.847)

27. Secondary Outcome: Main Study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Vitality Domain Score at Months 1, 6, 12, 18, 24, 30, and 36
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The 4-item measure of vitality captures a broad range of subjective evaluations of well-being from feelings of tiredness and being worn out to feeling full of energy all or most of the time. Norm-based domain scores were used in the analyses; each of which had a population mean of 50 with a SD of 10 points, and ranged from minus infinity to plus infinity. A higher vitality domain score represents better vitality.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | 5.92 (10.160)
  Change at Month 6: number analyzed (Participants) | 636
  Change at Month 6 | 6.03 (10.546)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | 6.72 (10.367)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | 6.67 (10.147)
  Change at Month 24: number analyzed (Participants) | 504
  Change at Month 24 | 7.10 (10.828)
  Change at Month 30: number analyzed (Participants) | 474
  Change at Month 30 | 7.62 (10.808)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | 7.65 (10.403)

28. Secondary Outcome: Main Study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Social Functioning Domain Score at Months 1, 6, 12, 18, 24, 30, and 36
Description: The SF-36v2 acute was a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The 2-item social functioning scale assessed health-related effects on quantity and quality of social activities. Norm-based domain scores were used in the analyses; each of which had a population mean of 50 with a SD of 10 points, and ranged from minus infinity to plus infinity. A higher social functioning domain score represented better social functioning.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | 6.08 (11.028)
  Change at Month 6: number analyzed (Participants) | 636
  Change at Month 6 | 6.51 (10.923)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | 7.16 (10.932)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | 6.76 (11.272)
  Change at Month 24: number analyzed (Participants) | 504
  Change at Month 24 | 7.28 (11.487)
  Change at Month 30: number analyzed (Participants) | 473
  Change at Month 30 | 7.64 (11.597)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | 7.83 (11.977)

29. Secondary Outcome: Main Study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2 ) Role-Emotional Domain Score at Months 1, 6, 12, 18, 24, 30, and 36
Description: The SF-36v2 acute was a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The 3-item role-emotional scale assessed mental health-related role limitations in terms of a) time spent in work or other usual activities; b) amount of work or activities accomplished; c) care with which work or other activities were performed. Norm-based domain scores were used in the analyses; each of which had a population mean of 50 with a SD of 10 points, and ranged from minus infinity to plus infinity. A higher role-emotional domain score represented better role-emotional functioning.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 668
  Change at Month 1 | 5.40 (11.962)
  Change at Month 6: number analyzed (Participants) | 632
  Change at Month 6 | 5.39 (12.445)
  Change at Month 12: number analyzed (Participants) | 578
  Change at Month 12 | 5.73 (12.235)
  Change at Month 18: number analyzed (Participants) | 534
  Change at Month 18 | 6.71 (12.647)
  Change at Month 24: number analyzed (Participants) | 502
  Change at Month 24 | 6.82 (12.154)
  Change at Month 30: number analyzed (Participants) | 473
  Change at Month 30 | 6.54 (12.843)
  Change at Month 36: number analyzed (Participants) | 384
  Change at Month 36 | 6.95 (12.859)

30. Secondary Outcome: Main Study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2 ) Mental Health Domain Score at Months 1, 6, 12, 18, 24, 30, and 36
Description: The SF-36v2 acute was a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The 5-item mental health scale includes 1 or more items from each of 4 major mental health dimensions: anxiety, depression, loss of behavioral/emotional control, and psychological well-being. Norm-based domain scores were used in the analyses; each of which had a population mean of 50 with a SD of 10 points, and ranged from minus infinity to plus infinity. A higher mental health domain score represented better mental health functioning.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | 4.85 (10.306)
  Change at Month 6: number analyzed (Participants) | 636
  Change at Month 6 | 5.39 (10.893)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | 5.56 (10.781)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | 5.82 (10.730)
  Change at Month 24: number analyzed (Participants) | 504
  Change at Month 24 | 6.09 (11.247)
  Change at Month 30: number analyzed (Participants) | 474
  Change at Month 30 | 6.18 (11.278)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | 6.37 (11.199)

31. Secondary Outcome: Main Study: Change From Baseline in EuroQol- 5D Health Questionnaire 3-Level (EQ-5D-3L) Mobility Domain at Months 1, 6, 12, 18, 24, 30 and 36
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions i.e. mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The status of each dimension had 3 possible responses (1 =no problem, 2 =some problem 3 =severe problems) in the relevant health dimension. Higher score indicated a worsening health condition. Data for change from baseline in EQ-5D-3L mobility domain score were reported in this outcome measure.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30 and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | -0.24 (0.529)
  Change at Month 6: number analyzed (Participants) | 635
  Change at Month 6 | -0.30 (0.540)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | -0.28 (0.511)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | -0.30 (0.538)
  Change at Month 24: number analyzed (Participants) | 505
  Change at Month 24 | -0.31 (0.545)
  Change at Month 30: number analyzed (Participants) | 474
  Change at Month 30 | -0.30 (0.526)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | -0.32 (0.555)

32. Secondary Outcome: Main Study: Change From Baseline in EuroQol-5D Health Questionnaire 3-Level (EQ-5D-3L) Self-Care Domain at Months 1, 6, 12, 18, 24, 30 and 36
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions i.e. mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The status of each dimension had 3 possible responses (1 =no problem, 2 =some problem 3 =severe problems) in the relevant health dimension. Higher score indicated a worsening health condition. Data for change from baseline in EQ-5D-3L self-care domain score were reported in this measure.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 673
  Change at Month 1 | -0.19 (0.547)
  Change at Month 6: number analyzed (Participants) | 633
  Change at Month 6 | -0.20 (0.530)
  Change at Month 12: number analyzed (Participants) | 581
  Change at Month 12 | -0.19 (0.532)
  Change at Month 18: number analyzed (Participants) | 535
  Change at Month 18 | -0.21 (0.522)
  Change at Month 24: number analyzed (Participants) | 503
  Change at Month 24 | -0.21 (0.534)
  Change at Month 30: number analyzed (Participants) | 473
  Change at Month 30 | -0.23 (0.533)
  Change at Month 36: number analyzed (Participants) | 385
  Change at Month 36 | -0.24 (0.589)

33. Secondary Outcome: Main Study: Change From Baseline in EuroQol-5D Health Questionnaire 3-Level (EQ-5D-3L) Usual Activities Domain at Months 1, 6, 12, 18, 24, 30 and 36
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions i.e. mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The status of each dimension had 3 possible responses (1 =no problem, 2 =some problem 3 =severe problems) in the relevant health dimension. Higher score indicated a worsening health condition. Data for change from baseline in EQ-5D-3L usual activities domain score were reported in this measure.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | -0.27 (0.588)
  Change at Month 6: number analyzed (Participants) | 635
  Change at Month 6 | -0.30 (0.539)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | -0.33 (0.547)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | -0.32 (0.579)
  Change at Month 24: number analyzed (Participants) | 505
  Change at Month 24 | -0.36 (0.547)
  Change at Month 30: number analyzed (Participants) | 474
  Change at Month 30 | -0.34 (0.571)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | -0.35 (0.594)

34. Secondary Outcome: Main Study: Change From Baseline in EuroQol-5D Health Questionnaire 3-Level (EQ-5D-3L) Pain/Discomfort Domain at Months 1, 6, 12, 18, 24, 30 and 36
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions i.e. mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The status of each dimension had 3 possible responses (1 =no problem, 2 =some problem 3 =severe problems) in the relevant health dimension. Higher score indicated a worsening health condition. Data for change from baseline in EQ-5D-3L pain/discomfort domain score were reported in this measure.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | -0.31 (0.557)
  Change at Month 6: number analyzed (Participants) | 635
  Change at Month 6 | -0.32 (0.570)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | -0.36 (0.568)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | -0.40 (0.584)
  Change at Month 24: number analyzed (Participants) | 505
  Change at Month 24 | -0.41 (0.602)
  Change at Month 30: number analyzed (Participants) | 474
  Change at Month 30 | -0.41 (0.601)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | -0.40 (0.613)

35. Secondary Outcome: Main Study: Change From Baseline in EuroQol-5D Health Questionnaire 3-Level (EQ-5D-3L) Anxiety/Depression Domain at Months 1, 6, 12, 18, 24, 30 and 36
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions i.e. mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The status of each dimension had 3 possible responses (1 =no problem, 2 =some problem 3 =severe problems) in the relevant health dimension. Higher score indicated a worsening health condition. Data for change from baseline in EQ-5D-3L anxiety/depression domain score were reported in this outcome measure.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | -0.23 (0.600)
  Change at Month 6: number analyzed (Participants) | 635
  Change at Month 6 | -0.26 (0.623)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | -0.25 (0.594)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | -0.26 (0.604)
  Change at Month 24: number analyzed (Participants) | 505
  Change at Month 24 | -0.29 (0.605)
  Change at Month 30: number analyzed (Participants) | 473
  Change at Month 30 | -0.31 (0.608)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | -0.29 (0.651)

36. Secondary Outcome: Main Study: Change From Baseline in EuroQol - Visual Analog Scale (EQ-VAS) Your Own Health State Today Domain at Months 1, 6, 12, 18, 24, 30 and 36
Description: The EQ VAS recorded the participant's self-rated health on a vertical VAS as standard vertical 0 (worst imaginable health state) to 100 mm (best imaginable health state) (similar to a thermometer) for recording an individual's rating for their current health-related quality of life state; higher score indicated a better health state.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
millimeter
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | 14.12 (24.928)
  Change at Month 6: number analyzed (Participants) | 636
  Change at Month 6 | 15.71 (25.871)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | 16.00 (24.896)
  Change at Month 18: number analyzed (Participants) | 535
  Change at Month 18 | 16.68 (24.746)
  Change at Month 24: number analyzed (Participants) | 505
  Change at Month 24 | 17.43 (25.226)
  Change at Month 30: number analyzed (Participants) | 473
  Change at Month 30 | 17.87 (25.363)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | 18.07 (25.185)

37. Secondary Outcome: Main Study: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Total Score at Months 1, 6, 12, 18, 24, 30 and 36
Description: FACIT-F:13-item questionnaire answered by participants,with each item scaled from 0(not at all) to 4(very much). 3 endpoints were derived:1)change in FACIT-F experience domain(score 0-20, higher score indicate less fatigue experience),calculated by summing 5 items(felt fatigued,felt weak all over,felt listless ["washed out"],felt tired,had energy; 2)change in FACIT-F impact domain(score 0-32,higher score indicate less fatigue impact on daily functioning),calculated by summing remaining 8 items(had trouble starting things as tired,had trouble finishing things as tired,was able to do usual activities,needed to sleep during day,too tired to eat,needed help doing my usual activities,frustrated by being too tired to do things wanted to do,had to limit my social activity because tired); 3)change in FACIT-F total score(0-52):calculated by summing 13 items,higher score indicated lower level of fatigue, better participant status. All responses were added with equal weight to get total score.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | 7.0 (9.78)
  Change at Month 6: number analyzed (Participants) | 636
  Change at Month 6 | 7.7 (10.13)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | 7.8 (9.70)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | 8.1 (10.06)
  Change at Month 24: number analyzed (Participants) | 506
  Change at Month 24 | 8.3 (10.61)
  Change at Month 30: number analyzed (Participants) | 474
  Change at Month 30 | 8.7 (10.93)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | 9.1 (11.05)

38. Secondary Outcome: Main Study: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Experience Domain Score at Months 1, 6, 12, 18, 24, 30 and 36
Description: FACIT-F:13-item questionnaire answered by participants,with each item scaled from 0(not at all) to 4(very much). 3 endpoints were derived:1)change in FACIT-F experience domain(score 0-20, higher score indicate less fatigue experience),calculated by summing 5 items(felt fatigued,felt weak all over,felt listless ["washed out"],felt tired,had energy; 2)change in FACIT-F impact domain(score 0-32,higher score indicate less fatigue impact on daily functioning),calculated by summing remaining 8 items(had trouble starting things as tired,had trouble finishing things as tired,was able to do usual activities,needed to sleep during day,too tired to eat,needed help doing my usual activities,frustrated by being too tired to do things wanted to do,had to limit my social activity because tired); 3)change in FACIT-F total score(0-52,higher score indicated lower level of fatigue, better participant status):calculated by summing 13 items, all responses were added with equal weight to get total score.
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | 3.1 (4.47)
  Change at Month 6: number analyzed (Participants) | 636
  Change at Month 6 | 3.4 (4.61)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | 3.5 (4.48)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | 3.6 (4.63)
  Change at Month 24: number analyzed (Participants) | 506
  Change at Month 24 | 3.7 (4.93)
  Change at Month 30: number analyzed (Participants) | 474
  Change at Month 30 | 3.9 (5.02)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | 4.0 (4.90)

39. Secondary Outcome: Main Study: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Impact Domain Score at Months 1, 6, 12, 18, 24, 30, and 36
Description: as for outcome 38
Time Frame: Main Study: Baseline (Day 1), Months 1, 6, 12, 18, 24, 30, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 686
units on a scale
  Change at Month 1: number analyzed (Participants) | 674
  Change at Month 1 | 3.9 (5.98)
  Change at Month 6: number analyzed (Participants) | 636
  Change at Month 6 | 4.2 (6.19)
  Change at Month 12: number analyzed (Participants) | 582
  Change at Month 12 | 4.4 (5.88)
  Change at Month 18: number analyzed (Participants) | 536
  Change at Month 18 | 4.5 (6.05)
  Change at Month 24: number analyzed (Participants) | 506
  Change at Month 24 | 4.6 (6.34)
  Change at Month 30: number analyzed (Participants) | 474
  Change at Month 30 | 4.8 (6.46)
  Change at Month 36: number analyzed (Participants) | 386
  Change at Month 36 | 5.0 (6.77)

40. Secondary Outcome: Sub-study: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Months 1, 3, 9 and 12
Description: HAQ-DI assessed the degree of difficulty a participant has experienced during the past week in 8 domains of daily living activities: dressing/grooming, arising, eating, walking, reach, grip, hygiene, and other activities. There were total of 2-3 items distributed in each of these 8 domains. Each item was scored for level of difficulty on a 4-point scale from 0 to 3: 0= no difficulty; 1= some difficulty; 2= much difficulty; 3= unable to do. Overall score was computed as the sum of domain score and divided by the number of domains answered. Total possible HAQ-DI score range 0 (least difficulty) and 3 (extreme difficulty), where higher score indicated more difficulty while performing daily living activities.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 9 and 12
Population: FAS for sub-study included all participants who were randomized to the sub-study and received at least 1 dose of (tofacitinib, MTX or placebo).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | -0.0164 (0.02438) | 0.0322 (0.02411)
  Change at Month 3 | 0.0057 (0.02512) | 0.0381 (0.02474)
  Change at Month 9 | 0.0720 (0.03195) | 0.0663 (0.03125)
  Change at Month 12 | 0.0467 (0.02998) | 0.0563 (0.02941)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: Change at Month 1: Results were based on a repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline value; a common unstructured covariance matrix was used; Test type: Other; LS Mean Difference = 0.0486, 95% CI 2-sided [-0.0192 to 0.1163]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: Change at Month 3: Results were based on a repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline value; a common unstructured covariance matrix was used; Test type: Other; LS Mean Difference = 0.0325, 95% CI 2-sided [-0.0372 to 0.1021]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: Change at Month 9: Results were based on a repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline value; a common unstructured covariance matrix was used; Test type: Other; LS Mean Difference = -0.0058, 95% CI 2-sided [-0.0941 to 0.0825]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: Change at Month 12: Results were based on a repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline value; a common unstructured covariance matrix was used; Test type: Other; LS Mean Difference = 0.0096, 95% CI 2-sided [-0.0734 to 0.0927]

41. Secondary Outcome: Sub-study: Change From Baseline in Psoriatic Arthritis Disease Activity Score (PASDAS) at Months 1, 3, 9 and 12
Description: PASDAS was composite PsA disease activity score that included following components: Physician and patient global assessment of disease activity (assessed on a 0-100 VAS) in mm, swollen (66 joints) and tender joint counts (68 joints), Leeds enthesitis index (enthesitis assessed at 6 sites; total score of 0-6), tender dactylitic digit score (scored on a scale of 0-3, where 0= no tenderness and 3= extreme tenderness), SF-36 physical component summary (norm-based domain score were used in analyses; with a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity) and CRP in mg/L. PASDAS was composite score and was a weighted index with score range of 0 to 10, where higher score indicated more severe disease.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 9 and 12
Population: as for outcome 40
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | 0.000 (0.0701) | 0.032 (0.0696)
  Change at Month 3 | 0.188 (0.0869) | 0.165 (0.0868)
  Change at Month 9 | 0.158 (0.0934) | 0.371 (0.0912)
  Change at Month 12 | 0.194 (0.0898) | 0.133 (0.0882)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS Mean Difference = 0.032, 95% CI 2-sided [-0.163 to 0.227]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS Mean Difference = -0.024, 95% CI 2-sided [-0.266 to 0.219]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS Mean Difference = 0.213, 95% CI 2-sided [-0.045 to 0.470]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS Mean Difference = -0.061, 95% CI 2-sided [-0.309 to 0.188]

42. Secondary Outcome: Sub-study: Percentage of Participants Achieving Psoriatic Arthritis Response Criteria (PsARC) at Months 1, 3, 6, 9 and 12
Description: PsARC was comprised of 4 clinical improvement criteria: >=20% improvement in PhyGA (VAS), >=20% improvement in PtGA; and >= 30% reduction in the number of tender joints; and >=30% reduction in the number of swollen joints. PtGA: participant assessed health on VAS, 0 mm (very well) to 100 mm (worst health condition), higher score = worse condition. PhyGA: physician judged participants' pain on VAS, 0 (no pain) to 100 mm (extreme pain), higher score = more pain. To achieve a clinical response, the participant must improve in 2 of the 4 PsARC criteria, 1 of which has to be the number of tender or swollen joints and none of the 4 score could worsen.
Time Frame: Months 1, 3, 6, 9 and 12
Population: FAS for sub-study included all participants who were randomized to the sub-study and received at least one dose of the sub-study drug (tofacitinib, MTX or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
percentage of participants
  Month 1 | 12.36 | 12.22
  Month 3 | 11.24 | 6.67
  Month 6 | 12.36 | 6.67
  Month 9 | 12.36 | 10.00
  Month 12 | 13.48 | 3.33
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: Month 1: Two-sided 95% CI was based on the normal approximation for the difference in binomial proportions; Test type: Other; Difference in percentage of participants = -0.14, 95% CI 2-sided [-9.76 to 9.48]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: Month 3: Two-sided 95% CI was based on the normal approximation for the difference in binomial proportions; Test type: Other; Difference in percentage of participants = -4.57, 95% CI 2-sided [-12.91 to 3.77]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: Month 6: Two-sided 95% CI was based on the normal approximation for the difference in binomial proportions; Test type: Other; Difference in percentage of participants = -5.69, 95% CI 2-sided [-14.26 to 2.87]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: Month 9: Two-sided 95% CI was based on the normal approximation for the difference in binomial proportions; Test type: Other; Difference in percentage of participants = -2.36, 95% CI 2-sided [-11.59 to 6.87]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: Month 12: Two-sided 95% CI was based on the normal approximation for the difference in binomial proportions; Test type: Other; Difference in percentage of participants = -10.15, 95% CI 2-sided [-18.16 to -2.14]

43. Secondary Outcome: Sub-study: Change From Baseline in Physician's Global Assessment of Psoriasis (PGA-PsO) Score (For Participants With Baseline PGA-PsO Score >0 ) at Months 1, 3, 6, 9 and 12
Description: The PGA-PsO is a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling were scored separately over the whole body according to a 5-point severity scale (0-4). Higher score indicated higher disease severity. Severity score for each erythema, induration and scaling were summed and averaged after which the total average was rounded to the nearest whole number score to determine a PGA-PsO score on a scale of 0 to 4 (0= clear, except for any residual discoloration, 1= almost clear, 2= mild, 3= moderate, 4= severe).
Time Frame: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: Analysis population included all participants who were randomized to the sub-study and received at least one dose of the sub-study drug (tofacitinib, MTX or placebo) with baseline PGA-PsO score>0.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 41 | 33
units on a scale
  Change at Month 1 | -0.1 (0.10) | 0.2 (0.11)
  Change at Month 3 | -0.1 (0.12) | 0.1 (0.14)
  Change at Month 6 | -0.1 (0.11) | 0.2 (0.12)
  Change at Month 9 | -0.3 (0.13) | 0.2 (0.13)
  Change at Month 12 | 0.0 (0.15) | 0.3 (0.15)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.2, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.2, 95% CI 2-sided [-0.1 to 0.6]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: Change at Month 6: Results were based on a repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline value; a common unstructured covariance matrix was used; Test type: Other; LS mean difference = 0.3, 95% CI 2-sided [0.0 to 0.6]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.5, 95% CI 2-sided [0.1 to 0.8]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]

44. Secondary Outcome: Sub-study: Percent Change From Baseline in Body Surface Area (BSA) (For Participants With BSA >0%) Psoriasis at Months 1, 3, 6, 9 and 12
Description: Assessment of BSA with psoriasis was estimated by means of the handprint method, where the full palmar hand of the participant (fully extended palm, fingers and thumb together) represented approximately 1% of the total BSA. Body regions are assigned specific number of handprints with percentage (Head and neck = 10 handprints [1 handprint =10%], upper extremities = 20 handprints [1 handprint =5%], Trunk (including axillae and groin) = 30 handprints [1 handprint =3.33%], lower extremities (including buttocks) = 40 handprints [1 handprint =2.5%]. The number of handprints of psoriatic skin in a body region was used to determine the extent (%) to which a body region was involved with psoriasis. The total BSA affected was the summation of individual regions affected.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: Analysis population included all participants who were randomized to the sub-study and received at least one dose of the sub-study drug (tofacitinib, MTX or placebo) with baseline BSA >0%. Here, "Number analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 47 | 42
percent change
  At Month 1: number analyzed (Participants) | 44 | 42
  At Month 1 | 28.47 (13.497) | 9.04 (13.972)
  At Month 3: number analyzed (Participants) | 44 | 41
  At Month 3 | 43.58 (18.679) | 13.47 (19.348)
  At Month 6: number analyzed (Participants) | 42 | 41
  At Month 6 | 41.51 (20.745) | 17.19 (21.157)
  At Month 9: number analyzed (Participants) | 40 | 40
  At Month 9 | 35.36 (17.309) | 23.72 (17.691)
  At Month 12: number analyzed (Participants) | 39 | 38
  At Month 12 | 34.74 (19.909) | 41.75 (20.333)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: At Month 1: Results were based on a repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline value; a common unstructured covariance matrix was used; Test type: Other; LS mean difference = -19.43, 95% CI 2-sided [-58.06 to 19.21]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: At Month 3: Results were based on a repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline value; a common unstructured covariance matrix was used; Test type: Other; LS mean difference = -30.11, 95% CI 2-sided [-83.58 to 23.37]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: At Month 6: Results were based on a repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline value; a common unstructured covariance matrix was used; Test type: Other; LS mean difference = -24.33, 95% CI 2-sided [-83.35 to 34.69]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: At Month 9: Results were based on a repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline value; a common unstructured covariance matrix was used; Test type: Other; LS mean difference = -11.64, 95% CI 2-sided [-60.87 to 37.58]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; Tofacitinib 5 mg BID + Placebo Vs Tofacitinib 5 mg BID +MTX: At Month 12: Results were based on a repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline value; a common unstructured covariance matrix was used; Test type: Other; LS mean difference = 7.02, 95% CI 2-sided [-49.73 to 63.77]

45. Secondary Outcome: Sub-study: Change From Baseline in Dactylitis Severity Score (DSS) (For Participants With Baseline DSS >0) at Months 1, 3, 6, 9 and 12
Description: Dactylitis was characterized by swelling of the entire finger or toe. The DSS was a function of finger circumference and tenderness, assessed and summed across all dactylitic digits. The severity of dactylitis was scored on a scale of 0-3, where 0 =no tenderness and 3 =extreme tenderness in each digit of the hands and feet. The range of total dactylitis score for a participant was 0-60. Higher score indicated greater degree of tenderness.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: Analysis population included all participants who were randomized to the sub-study and received at least one dose of the sub-study drug (tofacitinib, MTX or placebo) with baseline DSS >0. Here, "Number analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 7 | 1
units on a scale
  Change at Month 1 | -0.4 (0.79) | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Change at Month 3: number analyzed (Participants) | 6 | 1
  Change at Month 3 | -0.3 (0.52) | -1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Change at Month 6: number analyzed (Participants) | 6 | 1
  Change at Month 6 | -0.3 (0.52) | -1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Change at Month 9: number analyzed (Participants) | 6 | 1
  Change at Month 9 | -0.3 (0.52) | -1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Change at Month 12: number analyzed (Participants) | 6 | 1
  Change at Month 12 | -0.3 (0.52) | -1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

46. Secondary Outcome: Sub-study: Percentage of Participants With Absence of Dactylitis (For Participants With Baseline DSS >0) at Months 1, 3, 6, 9 and 12
Description: as for outcome 45
Time Frame: Sub-study: Months 1, 3, 6, 9 and 12
Population: Analysis population included all participants who were randomized to the sub-study and received at least one dose of the sub-study drug (tofacitinib, MTX or placebo) with baseline DSS >0.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 7 | 1
percentage of participants
  Month 1 | 14.29 | 0.0
  Month 3 | 14.29 | 0.0
  Month 6 | 14.29 | 0.0
  Month 9 | 14.29 | 0.0
  Month 12 | 14.29 | 0.0
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 1]; Test type: Other; Difference in percentage of participants = 6.25, 95% CI 2-sided [-59.58 to 72.08]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 2]; Test type: Other; Difference in percentage of participants = 6.25, 95% CI 2-sided [-59.58 to 72.08]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 3]; Test type: Other; Difference in percentage of participants = 6.25, 95% CI 2-sided [-59.58 to 72.08]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 4]; Test type: Other; Difference in percentage of participants = 6.25, 95% CI 2-sided [-59.58 to 72.08]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 5]; Test type: Other; Difference in percentage of participants = 6.25, 95% CI 2-sided [-59.58 to 72.08]

47. Secondary Outcome: Sub-study: Change From Baseline in Leeds Enthesitis Index (LEI) (For Participants With Baseline LEI >0) at Months 1, 3, 6, 9 and 12
Description: as for outcome 17
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: Analysis population included all participants who were randomized to the sub-study and received at least one dose of the sub-study drug (tofacitinib, MTX or placebo) and with baseline Leeds enthesitis index >0. Here, "Number analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 15 | 16
units on a scale
  Change at Month 1 | -0.2 (0.25) | -0.4 (0.24)
  Change at Month 3: number analyzed (Participants) | 15 | 15
  Change at Month 3 | -0.3 (0.23) | -0.5 (0.23)
  Change at Month 6 | -0.5 (0.29) | -0.7 (0.28)
  Change at Month 9 | -0.3 (0.29) | 0.0 (0.28)
  Change at Month 12: number analyzed (Participants) | 15 | 15
  Change at Month 12 | -0.5 (0.28) | -0.3 (0.27)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = -0.2, 95% CI 2-sided [-0.9 to 0.5]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = -0.2, 95% CI 2-sided [-0.9 to 0.5]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -0.2, 95% CI 2-sided [-1.1 to 0.6]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.2, 95% CI 2-sided [-0.6 to 1.1]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.2, 95% CI 2-sided [-0.6 to 1.0]

48. Secondary Outcome: Sub-study: Leeds Enthesitis Index (LEI) (For Participants With Baseline LEI =0) at Months 1, 3, 6, 9 and 12
Description: as for outcome 17
Time Frame: Sub-study: Months 1, 3, 6, 9 and 12
Population: Analysis population included all participants who were randomized to the sub-study and received at least one dose of the sub-study drug (tofacitinib, MTX or placebo) with baseline LEI =0. Here, "Number analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 74 | 74
units on a scale
  Month 1: number analyzed (Participants) | 72 | 73
  Month 1 | 0.2 (0.64) | 0.1 (0.58)
  Month 3: number analyzed (Participants) | 71 | 72
  Month 3 | 0.2 (0.56) | 0.0 (0.24)
  Month 6: number analyzed (Participants) | 69 | 72
  Month 6 | 0.2 (0.76) | 0.2 (0.82)
  Month 9: number analyzed (Participants) | 68 | 71
  Month 9 | 0.1 (0.24) | 0.1 (0.46)
  Month 12: number analyzed (Participants) | 68 | 70
  Month 12 | 0.2 (0.67) | 0.1 (0.49)

49. Secondary Outcome: Sub-study: Percentage of Participants With Absence of Enthesitis Assessed Using Leeds Enthesitis Index (LEI) (For Participants With Baseline LEI >0) at Months 1, 3, 6, 9 and 12
Description: as for outcome 17
Time Frame: Sub-study: Months 1, 3, 6, 9 and 12
Population: Analysis population included all participants who were randomized to the sub-study and received at least one dose of the sub-study drug (tofacitinib, MTX or placebo) with baseline LEI >0.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 15 | 16
percentage of participants
  Month 1 | 13.33 | 25.00
  Month 3 | 13.33 | 43.75
  Month 6 | 26.67 | 56.25
  Month 9 | 13.33 | 37.50
  Month 12 | 26.67 | 43.75
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 1]; Test type: Other; Difference in percentage of participants = 11.67, 95% CI 2-sided [-15.65 to 38.98]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 2]; Test type: Other; Difference in percentage of participants = 30.42, 95% CI 2-sided [0.64 to 60.20]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 3]; Test type: Other; Difference in percentage of participants = 29.58, 95% CI 2-sided [-3.46 to 62.62]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 4]; Test type: Other; Difference in percentage of participants = 24.17, 95% CI 2-sided [-5.14 to 53.47]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 5]; Test type: Other; Difference in percentage of participants = 17.08, 95% CI 2-sided [-15.96 to 50.12]

50. Secondary Outcome: Sub-study: Percentage of Participants With Minimal Disease Activity (MDA) at Months 1, 3, 6, 9 and 12
Description: A psoriatic arthritis participant was considered with minimal disease activity if participant had >= 5 of 7 criteria: 1) tender/painful joint count less than or equals to (<=) 1; (2) swollen joint count <=1; (3) BSA <=3%; (4) Patient Assessment of Arthritis Pain (VAS) <=15 mm; (5) PtGA (VAS) <=20 mm; (6) HAQ-DI score <=0.5; (7) tender entheseal points (using LEI) <=1.
Time Frame: Sub-study: Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
percentage of participants
  Month 1 | 50.56 | 55.56
  Month 3 | 50.56 | 54.44
  Month 6 | 46.07 | 48.89
  Month 9 | 42.70 | 46.67
  Month 12 | 41.57 | 44.44
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 1]; Test type: Other; Difference in percentage of participants = 4.99, 95% CI 2-sided [-9.61 to 19.60]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 2]; Test type: Other; Difference in percentage of participants = 3.88, 95% CI 2-sided [-10.74 to 18.50]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 3]; Test type: Other; Difference in percentage of participants = 2.82, 95% CI 2-sided [-11.80 to 17.45]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 4]; Test type: Other; Difference in percentage of participants = 3.97, 95% CI 2-sided [-10.58 to 18.52]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 42, analysis 5]; Test type: Other; Difference in percentage of participants = 2.87, 95% CI 2-sided [-11.63 to 17.37]

51. Secondary Outcome: Sub-study: Change From Baseline in Tender/Painful Joint Count at Months 1, 3, 6, 9 and 12
Description: 68 joints were assessed to determine joints that are considered tender or painful. Response to pressure/motion on each joint was assessed using the following scale: Present/Absent/Not Done/Done/Not Applicable (to be used for artificial or missing joints). The 68 joints assessed were: 1) Upper Body: temporomandibular, sternoclavicular, acromioclavicular. 2) Upper Extremity: shoulder, elbow, wrist (includes radiocarpal, carpal and carpometacarpal considered as one unit), metacarpophalangeals (MCP I, II, III, IV, V), thumb interphalangeal (IP), proximal interphalangeals (PIP II, III, IV, V), distal interphalangeals (DIP II, III, IV, V). 3) Lower Extremity: hip, knee, ankle, tarsus (includes subtalar, transverse tarsal and tarsometatarsal considered as one unit), metatarsophalangeals (MTP I, II, III, IV, V), great toe IP, proximal and distal interphalangeals combined (PIP II, III, IV, V).
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: tender/painful joints
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
tender/painful joints
  Change at Month 1 | 0.7 (0.37) | 0.3 (0.37)
  Change at Month 3 | 1.3 (0.44) | 0.9 (0.44)
  Change at Month 6 | 0.5 (0.37) | 0.5 (0.37)
  Change at Month 9 | 0.4 (0.33) | 0.4 (0.32)
  Change at Month 12 | 0.3 (0.32) | 0.5 (0.32)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = -0.4, 95% CI 2-sided [-1.5 to 0.6]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = -0.4, 95% CI 2-sided [-1.6 to 0.8]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-1.0 to 1.0]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.9 to 0.9]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.2, 95% CI 2-sided [-0.7 to 1.1]

52. Secondary Outcome: Sub-study: Change From Baseline in Swollen Joint Count at Months 1, 3, 6, 9 and 12
Description: Joints were assessed for swelling using the following scale: Present/Absent/Not Done/Not Applicable (to be used for artificial or missing joints). Sixty-six (66) joints were assessed for swelling. The 66 joints assessed were: 1) Upper Body: temporomandibular, sternoclavicular, acromioclavicular. 2) Upper Extremity: shoulder, elbow, wrist (includes radiocarpal, carpal and carpometacarpal considered as one unit), metacarpophalangeals (MCP I, II, III, IV, V), thumb interphalangeal (IP), proximal interphalangeals (PIP II, III, IV, V), distal interphalangeals (DIP II, III, IV, V). 3) Lower Extremity: knee, ankle, tarsus (includes subtalar, transverse tarsal and tarsometatarsal considered as one unit), metatarsophalangeals (MTP I, II, III, IV, V), great toe IP, proximal and distal interphalangeals combined (PIP II, III, IV, V).
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: swollen joints
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
swollen joints
  Change at Month 1 | -0.1 (0.14) | 0.0 (0.14)
  Change at Month 3 | 0.3 (0.21) | 0.3 (0.21)
  Change at Month 6 | 0.1 (0.16) | 0.1 (0.15)
  Change at Month 9 | 0.0 (0.17) | 0.2 (0.17)
  Change at Month 12 | 0.1 (0.14) | 0.0 (0.14)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [-0.3 to 0.5]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.6 to 0.6]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.4 to 0.5]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.2, 95% CI 2-sided [-0.3 to 0.7]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = -0.1, 95% CI 2-sided [-0.5 to 0.3]

53. Secondary Outcome: Sub-study: Change From Baseline in Physician's Global Assessment of Arthritis (PhyGA) at Months 1, 3, 6, 9 and 12
Description: The investigator or qualified assessor assessed how the participant's overall arthritis appeared at the time of the visit. This was an evaluation based on the participant's disease signs, functional capacity and physical examination, and independent of the PtGA and Patient Assessment of Arthritis Pain. The investigator's response was recorded using a 100 mm VAS where 0 =PSA not active at all and 100 =PSA extremely active. Higher score indicated more PSA.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
millimeter
  Change at Month 1 | -0.42 (0.992) | -0.17 (0.981)
  Change at Month 3 | 1.98 (1.225) | 2.76 (1.216)
  Change at Month 6 | 1.18 (0.983) | 1.65 (0.966)
  Change at Month 9 | 1.18 (1.316) | 3.35 (1.287)
  Change at Month 12 | 0.86 (1.127) | 0.75 (1.111)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.26, 95% CI 2-sided [-2.51 to 3.02]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.77, 95% CI 2-sided [-2.64 to 4.18]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = 0.47, 95% CI 2-sided [-2.26 to 3.20]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 2.18, 95% CI 2-sided [-1.46 to 5.81]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = -0.12, 95% CI 2-sided [-3.25 to 3.01]

54. Secondary Outcome: Sub-study: Change From Baseline in Patient's Global Assessment of Arthritis (PtGA) at Months 1, 3, 6, 9 and 12
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participant's response were recorded using a 0 - 100 mm VAS where 0 =not affected at all and 100 =extremely affected. Higher score indicated worse condition due to PSA.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
millimeter
  Change at Month 1 | 1.35 (1.277) | -0.68 (1.264)
  Change at Month 3 | 2.11 (1.537) | 1.68 (1.516)
  Change at Month 6 | 3.17 (1.725) | 4.45 (1.690)
  Change at Month 9 | 2.63 (1.691) | 3.27 (1.655)
  Change at Month 12 | 2.77 (1.629) | 2.65 (1.602)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = -2.03, 95% CI 2-sided [-5.58 to 1.52]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = -0.43, 95% CI 2-sided [-4.69 to 3.84]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = 1.29, 95% CI 2-sided [-3.48 to 6.06]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.64, 95% CI 2-sided [-4.03 to 5.32]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = -0.13, 95% CI 2-sided [-4.64 to 4.38]

55. Secondary Outcome: Sub-study: Change From Baseline in Patient's Assessment of Arthritis Pain at Months 1, 3, 6, 9 and 12
Description: Participants assessed the severity of their arthritis pain using a 100 mm VAS by placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponded to the magnitude of their pain. Higher score indicated more severe pain.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
millimeter
  Change at Month 1 | -0.05 (1.383) | -1.16 (1.370)
  Change at Month 3 | 1.59 (1.394) | 0.36 (1.380)
  Change at Month 6 | 3.12 (1.709) | 4.07 (1.674)
  Change at Month 9 | 2.44 (1.780) | 4.45 (1.741)
  Change at Month 12 | 2.69 (1.692) | 3.35 (1.664)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = -1.11, 95% CI 2-sided [-4.96 to 2.74]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = -1.23, 95% CI 2-sided [-5.11 to 2.65]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = 0.95, 95% CI 2-sided [-3.78 to 5.69]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 2.01, 95% CI 2-sided [-2.92 to 6.93]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.66, 95% CI 2-sided [-4.03 to 5.35]

56. Secondary Outcome: Sub-study: Change From Baseline in C-Reactive Protein (CRP) at Months 1, 3, 6, 9 and 12
Description: The test for CRP was a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
mg/L
  Change at Month 1 | -0.1171 (0.71654) | -0.2706 (0.70892)
  Change at Month 3 | -0.3625 (0.48088) | -0.9285 (0.47675)
  Change at Month 6 | 0.5354 (0.79954) | -0.2637 (0.78002)
  Change at Month 9 | -0.3217 (0.59271) | -0.2591 (0.57983)
  Change at Month 12 | -0.1005 (0.78650) | 0.2667 (0.77230)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = -0.1535, 95% CI 2-sided [-2.1444 to 1.8374]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = -0.5660, 95% CI 2-sided [-1.9054 to 0.7735]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -0.7991, 95% CI 2-sided [-3.0053 to 1.4071]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.0626, 95% CI 2-sided [-1.5767 to 1.7018]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.3672, 95% CI 2-sided [-1.8107 to 2.5450]

57. Secondary Outcome: Sub-study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Physical Component Summary Score at Months 1, 3, 6, 9 and 12
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. An additional item measures health transition. The 8 health domains are aggregated into two summary scores known as the PCS score and MCS score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a standard deviation (SD) of 10 points, and ranges from minus infinity to plus infinity. A higher PCS score represents better physical health status.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | -0.55 (0.424) | -0.22 (0.419)
  Change at Month 3 | -0.90 (0.492) | -0.57 (0.487)
  Change at Month 6 | -0.65 (0.480) | -1.42 (0.466)
  Change at Month 9 | -1.09 (0.607) | -1.85 (0.593)
  Change at Month 12 | -1.52 (0.533) | -1.00 (0.523)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.33, 95% CI 2-sided [-0.85 to 1.51]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.33, 95% CI 2-sided [-1.04 to 1.69]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -0.77, 95% CI 2-sided [-2.09 to 0.55]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = -0.77, 95% CI 2-sided [-2.44 to 0.91]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.52, 95% CI 2-sided [-0.96 to 2.00]

58. Secondary Outcome: Sub-study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Mental Component Summary Score at Months 1, 3, 6, 9 and 12
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. An additional item measures health transition. The 8 health domains are aggregated into two summary scores known as the PCS score and the MCS score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher MCS score represents better mental health status.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | 0.35 (0.630) | -0.11 (0.622)
  Change at Month 3 | 0.09 (0.642) | -0.77 (0.634)
  Change at Month 6 | -0.23 (0.733) | -0.89 (0.713)
  Change at Month 9 | -0.71 (0.749) | 0.06 (0.731)
  Change at Month 12 | -0.38 (0.694) | -0.47 (0.681)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = -0.47, 95% CI 2-sided [-2.22 to 1.29]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = -0.86, 95% CI 2-sided [-2.65 to 0.92]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -0.66, 95% CI 2-sided [-2.68 to 1.36]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.76, 95% CI 2-sided [-1.31 to 2.83]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = -0.09, 95% CI 2-sided [-2.01 to 1.84]

59. Secondary Outcome: Sub-study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Physical Functioning Domain Score at Months 1, 3, 6, 9 and 12
Description: SF-36v2 was a 36-item measure evaluating 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health. The 10 items of the physical functioning scale represented levels and kinds of limitations between extremes of physical activities, including lifting & carrying groceries; climbing stairs; bending, kneeling, or stooping; walking moderate distances; self-care limitations. The physical functioning items capture the presence & extent of physical limitations using a 3-level response continuum. Norm-based domain scores were used in the analyses; each of which had a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher physical functioning domain score represented better physical functioning.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | -0.37 (0.472) | -0.15 (0.467)
  Change at Month 3 | -0.50 (0.562) | -0.33 (0.556)
  Change at Month 6 | -0.27 (0.586) | -0.80 (0.571)
  Change at Month 9 | -1.43 (0.657) | -1.11 (0.643)
  Change at Month 12 | -1.01 (0.676) | -1.02 (0.664)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.22, 95% CI 2-sided [-1.09 to 1.53]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.17, 95% CI 2-sided [-1.39 to 1.73]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -0.53, 95% CI 2-sided [-2.15 to 1.08]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.32, 95% CI 2-sided [-1.49 to 2.13]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = -0.01, 95% CI 2-sided [-1.89 to 1.86]

60. Secondary Outcome: Sub-study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Role Physical Domain Score at Months 1, 3, 6, 9 and 12
Description: as for outcome 24
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | -0.27 (0.561) | 0.22 (0.555)
  Change at Month 3 | -1.04 (0.626) | 0.21 (0.619)
  Change at Month 6 | -1.57 (0.585) | -0.87 (0.569)
  Change at Month 9 | -0.64 (0.638) | -0.44 (0.624)
  Change at Month 12 | -1.85 (0.646) | -0.12 (0.635)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.48, 95% CI 2-sided [-1.08 to 2.05]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 1.25, 95% CI 2-sided [-0.49 to 2.99]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = 0.70, 95% CI 2-sided [-0.91 to 2.31]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.20, 95% CI 2-sided [-1.57 to 1.96]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 1.73, 95% CI 2-sided [-0.06 to 3.52]

61. Secondary Outcome: Sub-study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Bodily Pain Domain Score at Months 1, 3, 6, 9 and 12
Description: as for outcome 25
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | -0.77 (0.617) | -0.06 (0.609)
  Change at Month 3 | -1.59 (0.661) | -1.24 (0.652)
  Change at Month 6 | -0.61 (0.686) | -2.42 (0.669)
  Change at Month 9 | -1.29 (0.808) | -3.05 (0.790)
  Change at Month 12 | -1.69 (0.719) | -1.99 (0.706)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.71, 95% CI 2-sided [-1.01 to 2.42]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.34, 95% CI 2-sided [-1.49 to 2.18]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -1.81, 95% CI 2-sided [-3.70 to 0.09]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = -1.76, 95% CI 2-sided [-3.99 to 0.48]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = -0.30, 95% CI 2-sided [-2.30 to 1.69]

62. Secondary Outcome: Sub-study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) General Health Domain Score at Months 1, 3, 6, 9 and 12
Description: as for outcome 26
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | 0.20 (0.492) | -0.48 (0.487)
  Change at Month 3 | 0.34 (0.516) | -0.79 (0.511)
  Change at Month 6 | 0.24 (0.493) | -0.57 (0.481)
  Change at Month 9 | -0.48 (0.562) | -0.46 (0.551)
  Change at Month 12 | -0.32 (0.539) | -0.29 (0.530)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = -0.68, 95% CI 2-sided [-2.05 to 0.69]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = -1.13, 95% CI 2-sided [-2.57 to 0.31]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -0.81, 95% CI 2-sided [-2.17 to 0.56]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.01, 95% CI 2-sided [-1.54 to 1.57]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.04, 95% CI 2-sided [-1.46 to 1.53]

63. Secondary Outcome: Sub-study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Vitality Domain Score at Months 1, 3, 6, 9 and 12
Description: The SF-36v2 acute was a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The 4-item measure of vitality captures a broad range of subjective evaluations of well-being from feelings of tiredness and being worn out to feeling full of energy all or most of the time. Norm-based domain scores were used in the analyses; each of which had a population mean of 50 with a SD of 10 points, and ranged from minus infinity to plus infinity. A higher vitality domain score represented better vitality.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | -0.04 (0.614) | -0.39 (0.607)
  Change at Month 3 | -0.26 (0.593) | -1.12 (0.586)
  Change at Month 6 | 0.01 (0.705) | -1.70 (0.687)
  Change at Month 9 | -0.80 (0.645) | -1.27 (0.632)
  Change at Month 12 | -1.04 (0.640) | -0.09 (0.629)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = -0.36, 95% CI 2-sided [-2.06 to 1.35]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = -0.86, 95% CI 2-sided [-2.51 to 0.79]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -1.71, 95% CI 2-sided [-3.66 to 0.23]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = -0.47, 95% CI 2-sided [-2.25 to 1.32]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.95, 95% CI 2-sided [-0.82 to 2.73]

64. Secondary Outcome: Sub-study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Social Functioning Domain Score at Months 1, 3, 6, 9 and 12
Description: as for outcome 28
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | -0.99 (0.734) | -0.22 (0.726)
  Change at Month 3 | -0.80 (0.750) | -1.18 (0.740)
  Change at Month 6 | -1.16 (0.776) | -1.74 (0.757)
  Change at Month 9 | -1.50 (0.753) | -1.22 (0.737)
  Change at Month 12 | -1.81 (0.758) | -1.28 (0.746)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.78, 95% CI 2-sided [-1.27 to 2.82]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = -0.38, 95% CI 2-sided [-2.46 to 1.71]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -0.57, 95% CI 2-sided [-2.72 to 1.57]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.28, 95% CI 2-sided [-1.81 to 2.36]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.53, 95% CI 2-sided [-1.58 to 2.63]

65. Secondary Outcome: Sub-study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Role Emotional Domain Score at Months 1, 3, 6, 9 and 12
Description: as for outcome 29
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | 1.14 (0.716) | -0.53 (0.707)
  Change at Month 3 | 0.24 (0.807) | -0.38 (0.797)
  Change at Month 6 | -0.72 (0.788) | -0.82 (0.769)
  Change at Month 9 | -0.78 (0.803) | -0.06 (0.782)
  Change at Month 12 | -0.33 (0.835) | -1.11 (0.820)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = -1.67, 95% CI 2-sided [-3.67 to 0.32]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = -0.61, 95% CI 2-sided [-2.86 to 1.63]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -0.09, 95% CI 2-sided [-2.27 to 2.09]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.73, 95% CI 2-sided [-1.49 to 2.95]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = -0.79, 95% CI 2-sided [-3.10 to 1.53]

66. Secondary Outcome: Sub Study: Change From Baseline in Short-Form-36 Health Survey Version 2 (SF-36v2) Mental Health Domain Score at Months 1, 3, 6, 9 and 12
Description: as for outcome 30
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | -0.30 (0.676) | 0.63 (0.669)
  Change at Month 3 | -0.42 (0.661) | -0.31 (0.653)
  Change at Month 6 | -0.01 (0.780) | -0.26 (0.762)
  Change at Month 9 | -0.72 (0.724) | 0.35 (0.710)
  Change at Month 12 | -0.37 (0.723) | 0.01 (0.711)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.93, 95% CI 2-sided [-0.95 to 2.81]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.11, 95% CI 2-sided [-1.72 to 1.95]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -0.25, 95% CI 2-sided [-2.40 to 1.90]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 1.07, 95% CI 2-sided [-0.93 to 3.07]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.38, 95% CI 2-sided [-1.62 to 2.38]

67. Secondary Outcome: Sub Study: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Total Score at Months 1, 3, 6, 9 and 12
Description: as for outcome 37
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | -1.9 (0.61) | -1.1 (0.61)
  Change at Month 3 | -1.8 (0.59) | -1.3 (0.58)
  Change at Month 6 | -1.3 (0.61) | -2.0 (0.60)
  Change at Month 9 | -2.1 (0.65) | -1.0 (0.64)
  Change at Month 12 | -1.4 (0.66) | -0.7 (0.64)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.8, 95% CI 2-sided [-0.9 to 2.5]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.5, 95% CI 2-sided [-1.1 to 2.2]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -0.7, 95% CI 2-sided [-2.4 to 1.0]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 1.1, 95% CI 2-sided [-0.8 to 2.9]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.8, 95% CI 2-sided [-1.1 to 2.6]

68. Secondary Outcome: Sub Study: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Experience Domain Score at Months 1, 3, 6, 9 and 12
Description: as for outcome 38
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | -0.9 (0.29) | -0.5 (0.29)
  Change at Month 3 | -0.8 (0.31) | -0.9 (0.30)
  Change at Month 6 | -0.5 (0.29) | -1.3 (0.28)
  Change at Month 9 | -0.7 (0.31) | -0.8 (0.30)
  Change at Month 12 | -0.5 (0.31) | -0.5 (0.31)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.4, 95% CI 2-sided [-0.4 to 1.2]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = -0.1, 95% CI 2-sided [-1.0 to 0.7]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -0.7, 95% CI 2-sided [-1.6 to 0.1]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.9 to 0.8]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.9 to 0.8]

69. Secondary Outcome: Sub Study: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Impact Domain Score at Months 1, 3, 6, 9 and 12
Description: as for outcome 38
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | -1.1 (0.39) | -0.6 (0.39)
  Change at Month 3 | -1.1 (0.35) | -0.4 (0.35)
  Change at Month 6 | -0.8 (0.41) | -0.7 (0.40)
  Change at Month 9 | -1.4 (0.42) | -0.2 (0.41)
  Change at Month 12 | -0.9 (0.40) | -0.1 (0.40)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.5, 95% CI 2-sided [-0.6 to 1.6]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.7, 95% CI 2-sided [-0.3 to 1.7]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [-1.0 to 1.2]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 1.2, 95% CI 2-sided [0.0 to 2.3]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.8, 95% CI 2-sided [-0.3 to 1.9]

70. Secondary Outcome: Sub Study: Change From Baseline in EuroQol-5D Health Questionnaire 3-Level (EQ-5D-3L) Mobility Domain at Months 1, 3, 6, 9 and 12
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions i.e. mobility, self-care, usual activities, pain/discomfort and anxiety/depression) are assessed. The status of each dimension had 3 possible responses (1 =no problem, 2= some problem 3 =severe problems) in the relevant health dimension. Higher score indicated a worsening health condition. Data for change from baseline in EQ-5D-3L mobility domain score were reported in this measure.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | 0.0 (0.04) | 0.0 (0.04)
  Change at Month 3 | 0.0 (0.04) | 0.0 (0.04)
  Change at Month 6 | 0.0 (0.04) | 0.1 (0.04)
  Change at Month 9 | 0.0 (0.04) | 0.1 (0.04)
  Change at Month 12 | 0.0 (0.04) | 0.1 (0.04)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [0.0 to 0.2]

71. Secondary Outcome: Sub Study: Change From Baseline in EuroQol-5D Health Questionnaire 3-Level (EQ-5D-3L) Self-Care Domain at Months 1, 3, 6, 9 and 12
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions i.e. mobility, self-care, usual activities, pain/discomfort and anxiety/depression) are assessed. The status of each dimension had 3 possible responses (1 =no problem, 2= some problem 3 =severe problems) in the relevant health dimension. Higher score indicated a worsening health condition. Data for change from baseline in EQ-5D-3L self-care domain score were reported in this measure.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | 0.0 (0.03) | 0.0 (0.03)
  Change at Month 3 | 0.0 (0.03) | 0.0 (0.03)
  Change at Month 6 | 0.0 (0.04) | 0.0 (0.03)
  Change at Month 9 | 0.0 (0.04) | 0.0 (0.04)
  Change at Month 12 | 0.0 (0.04) | 0.1 (0.04)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [0.0 to 0.1]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [0.0 to 0.2]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [0.0 to 0.2]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.1]

72. Secondary Outcome: Sub Study: Change From Baseline in EuroQol-5D Health Questionnaire 3-Level (EQ-5D-3L) Usual Activities Domain at Months 1, 3, 6, 9 and 12
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions i.e. mobility, self-care, usual activities, pain/discomfort and anxiety/depression) are assessed. The status of each dimension had 3 possible responses (1 =no problem, 2= some problem 3 =severe problems) in the relevant health dimension. Higher score indicated a worsening health condition. Data for change from baseline in EQ-5D-3L usual activities domain score were reported in this measure.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | 0.0 (0.04) | 0.0 (0.04)
  Change at Month 3 | 0.0 (0.04) | 0.0 (0.04)
  Change at Month 6 | 0.0 (0.04) | 0.1 (0.04)
  Change at Month 9 | 0.1 (0.04) | 0.1 (0.04)
  Change at Month 12 | 0.0 (0.04) | 0.0 (0.04)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [0.0 to 0.2]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [-0.1 to 0.2]

73. Secondary Outcome: Sub Study: Change From Baseline in EuroQol-5D Health Questionnaire 3-Level (EQ-5D-3L) Pain/Discomfort Domain
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions i.e. mobility, self-care, usual activities, pain/discomfort and anxiety/depression) are assessed. The status of each dimension had 3 possible responses (1 =no problem, 2= some problem 3 =severe problems) in the relevant health dimension. Higher score indicated a worsening health condition. Data for change from baseline in EQ-5D-3L pain/discomfort domain score were reported in this measure.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | 0.1 (0.04) | 0.0 (0.04)
  Change at Month 3 | 0.1 (0.04) | 0.1 (0.04)
  Change at Month 6 | 0.1 (0.04) | 0.1 (0.04)
  Change at Month 9 | 0.1 (0.05) | 0.1 (0.05)
  Change at Month 12 | 0.1 (0.05) | 0.2 (0.05)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = 0.1, 95% CI 2-sided [-0.1 to 0.2]

74. Secondary Outcome: Sub Study: Change From Baseline in EuroQol-5D Health Questionnaire 3-Level (EQ-5D-3L) Anxiety/Depression Domain at Months 1, 3, 6, 9 and 12
Description: EQ-5D-3L, a health profile questionnaire was used to assess quality of life along 5 dimensions i.e. mobility, self-care, usual activities, pain/discomfort and anxiety/depression) are assessed. The status of each dimension had 3 possible responses (1 =no problem, 2= some problem 3 =severe problems) in the relevant health dimension. Higher score indicated a worsening health condition. Data for change from baseline in EQ-5D-3L anxiety/depression domain score were reported in this measure.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
units on a scale
  Change at Month 1 | 0.1 (0.04) | 0.0 (0.04)
  Change at Month 3 | 0.0 (0.05) | 0.0 (0.04)
  Change at Month 6 | 0.1 (0.05) | 0.0 (0.05)
  Change at Month 9 | 0.1 (0.05) | 0.0 (0.05)
  Change at Month 12 | 0.1 (0.05) | 0.0 (0.05)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = 0.0, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -0.1, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = -0.1, 95% CI 2-sided [-0.3 to 0.0]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = -0.1, 95% CI 2-sided [-0.2 to 0.0]

75. Secondary Outcome: Sub Study: Change From Baseline in EuroQol - Visual Analog Scale (EQ-VAS) Your Own Health State Today Domain at Months 1, 3, 6, 9 and 12
Description: The EQ VAS recorded the participant's self-rated health on a vertical VAS as standard verticle 0 (worst imaginable health state) to 100 mm (best imaginable health state) (similar to a thermometer) for recording an individual's rating for their current health-related quality of life state; higher score indicated a better health state.
Time Frame: Sub-study: Baseline (Day 1), Months 1, 3, 6, 9 and 12
Population: as for outcome 42
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
Number analyzed (Participants) | 89 | 90
millimeter
  Change at Month 1 | 2.0 (1.19) | -0.9 (1.16)
  Change at Month 3 | 0.5 (1.54) | -1.1 (1.52)
  Change at Month 6 | 4.4 (1.41) | -1.9 (1.38)
  Change at Month 9 | 2.5 (1.59) | -0.4 (1.56)
  Change at Month 12 | 3.0 (1.82) | -1.9 (1.78)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 1]; Test type: Other; LS mean difference = -2.9, 95% CI 2-sided [-6.2 to 0.4]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 2]; Test type: Other; LS mean difference = -1.5, 95% CI 2-sided [-5.8 to 2.7]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 43, analysis 3]; Test type: Other; LS mean difference = -6.3, 95% CI 2-sided [-10.2 to -2.4]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 3]; Test type: Other; LS mean difference = -2.8, 95% CI 2-sided [-7.3 to 1.6]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID + Methotrexate (MTX) vs Tofacitinib 5 mg BID + Placebo; [analysis description as in outcome 40, analysis 4]; Test type: Other; LS mean difference = -4.9, 95% CI 2-sided [-9.9 to 0.2]

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to last dose of main study (maximum up to 36 months) if not enrolled into sub-study or from baseline up to last dose of sub-study (maximum up to 48 months) if enrolled into sub-study
Description: Analysis performed on safety analysis set. As pre-specified in protocol/SAP, safety data were planned to be assessed as a single group (without regard to tofacitinib doses) in the main study. For the main study report, the analysis of the safety data included cumulative safety data from both the main and the sub-study as a single group. In addition, the safety data collected in the sub-study was analyzed for tofacitinib 5 mg BID + MTX and tofacitinib 5 mg BID + placebo, separately.
Groups:
- All Tofacitinib: Main Study: Participants with active PsA received tofacitinib 5 mg oral tablet, BID with or without allowed concomitant DMARDs examples as methotrexate, leflunomide or sulfasalazine, as background therapy, for up to 36 months. Tofacitinib dose was increased to 10 mg BID or decreased back to 5 mg BID per investigator's discretion. Sub-study: Participants from main study received tofacitinib 5 mg oral tablet BID with MTX capsules orally (dose range from 7.5 to 20 mg per week) or tofacitinib 5 mg oral tablet BID with MTX matched placebo capsules, for up to 12 months.
Arm/Group | All Tofacitinib | Tofacitinib 5 mg BID + Methotrexate (MTX) | Tofacitinib 5 mg BID + Placebo
All-Cause Mortality (participants affected / at risk) | 6/686 | 0/89 | 0/90
Serious Adverse Events (participants affected / at risk) | 115/686 | 3/89 | 4/90
Other Adverse Events (participants affected / at risk) | 457/686 | 25/89 | 24/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Tofacitinib (N=686) | Tofacitinib 5 mg BID + Methotrexate (MTX) (N=89) | Tofacitinib 5 mg BID + Placebo (N=90)
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 3 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Chorioretinopathy (Eye disorders) | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 2 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Nodule (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Epiglottitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
HIV infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Neurosyphilis (Infections and infestations) | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Pyoderma (Infections and infestations) | 1 | 0 | 0
Serratia sepsis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Heart rate decreased (Investigations) | 1 | 0 | 0
Cardiometabolic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Device loosening (Product Issues) | 1 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Breast disorder female (Reproductive system and breast disorders) | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Pneumonia herpes viral (Infections and infestations) | 1 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Vertebral lateral recess stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Miscarriage of partner (Social circumstances) | 1 | 0 | 0
Post thrombotic syndrome (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Tofacitinib (N=686) | Tofacitinib 5 mg BID + Methotrexate (MTX) (N=89) | Tofacitinib 5 mg BID + Placebo (N=90)
Anaemia (Blood and lymphatic system disorders) | 15 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 25 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 17 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 15 | 2 | 0
Nausea (Gastrointestinal disorders) | 27 | 0 | 0
Oedema peripheral (General disorders) | 14 | 0 | 0
Bronchitis (Infections and infestations) | 67 | 2 | 3
Gastroenteritis (Infections and infestations) | 19 | 0 | 0
Nasopharyngitis (Infections and infestations) | 104 | 1 | 3
Pharyngitis (Infections and infestations) | 38 | 3 | 3
Respiratory tract infection (Infections and infestations) | 17 | 0 | 0
Sinusitis (Infections and infestations) | 33 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 124 | 6 | 4
Urinary tract infection (Infections and infestations) | 66 | 3 | 4
Herpes zoster (Infections and infestations) | 26 | 2 | 1
Influenza (Infections and infestations) | 19 | 0 | 0
Oral herpes (Infections and infestations) | 19 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 24 | 0 | 0
Alanine aminotransferase increased (Investigations) | 34 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 21 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 36 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 22 | 0 | 0
Hepatic enzyme increased (Investigations) | 15 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 14 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 44 | 3 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 20 | 0 | 0
Headache (Nervous system disorders) | 32 | 2 | 0
Sciatica (Nervous system disorders) | 19 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 32 | 2 | 1
Hypertension (Vascular disorders) | 50 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT01976364/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT01976364/SAP_001.pdf